CLINICAL TRIAL: NCT02310568
Title: An 8-week, Randomized, Phase 2, Double-blind, Sequential Parallel-group Comparison Study Of Two Dose Levels Of Pf 06372865 Compared To Placebo As An Adjunctive Treatment In Outpatients With Inadequate Response To Standard Of Care For Generalized Anxiety Disorder
Brief Title: POC Study in Partially Responsive Generalized Anxiety Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study recruitment was terminated on 24 June 2015, due to a Pfizer business decision. This study was not terminated for reasons of safety or efficacy
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B7431007
Record Dates: First submitted 2014-10-24; First posted 2014-12-08 (Estimated); Results first posted 2016-11-15 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-09

CONDITIONS: Generalized Anxiety Disorder
Keywords: PF 06372865; generalized anxiety disorder; outpatient; safety; efficacy; suboptimal response
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — PF-06372865

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- PF 06372865 2.5 mg BID then placebo. (Experimental): PF 06372865 2.5 mg tablet 2 times daily for 4 weeks (Stage 1), followed by placebo 2 times daily for 4 weeks (Stage 2).
  Interventions: Drug: PF-06372865.
- PF 06372865 7.5 mg BID then placebo. (Experimental): PF 06372865 2.5 mg tablet 2 times daily for one week, then PF 06372865 7.5 mg tablet 2 times daily for 3 weeks (Stage 1), followed by placebo (2 times daily) for 4 weeks (Stage 2).
  Interventions: Drug: PF-06372865.
- Placebo then PF 06372865 2.5 mg BID. (Experimental): Placebo 2 times daily for 4 weeks (Stage 1), followed by PF 06372865 2.5 mg tablet 2 times daily for 4 weeks
  Interventions: Drug: PF-06372865.
- Placebo then PF 06372865 7.5 mg BID. (Experimental): Placebo 2 times daily for 4 weeks (Stage 1), followed by PF 06372865 2.5 mg tablet 2 times daily for one week, then PF 06372865 7.5 mg tablet 2 times daily for 3 weeks (Stage 2).
  Interventions: Drug: PF-06372865.
- Placebo followed by placebo. (Placebo Comparator): Placebo 2 times daily for 4 weeks (Stage 1) followed by Placebo 2 times daily for 4 weeks (Stage 2).
  Interventions: Drug: PF-06372865.

INTERVENTIONS:
Drug: PF-06372865. — Blinded PF 06372865 and matching placebo will be provided as tablets for oral administration.

SUMMARY:
This study aims to evaluate whether PF-06372865 is safe and effective in the treatment of sub-optimally controlled symptoms of generalized anxiety disorder during two 4-week treatment periods using a Sequential Parallel Comparison Design (SPCD). The study will use the Hamilton Anxiety Rating Scale (HAM-A) to measure change in symptoms from baseline for two doses of PF-06372865 compared to placebo.

ELIGIBILITY:
Inclusion criteria:

1. Outpatient males and females 18 65 years of age (inclusive).
2. Diagnostic and Statistical Manual of Mental Disorders Fourth edition Text Revised (DSM IV TR) diagnosis of GAD (DSM IV TR, 300.02), confirmed as primary diagnosis by the Mini international neuropsychiatric interview (MINI) structured interview.
3. All subjects must have a total HAM A (via SIGH A) score 22 at screening. In addition, scores at the baseline visit must also be within 20% of scores at screening.
4. Subjects must also have a Covi Anxiety Scale score of 9 and a Raskin Depression Scale score 7 at the Screening (Visit 1) visit to ensure predominance of anxiety symptoms over depression symptoms.
5. Taking an FDA approved GAD treatment (escitalopram 10 to 20 mg total daily dose, paroxetine 20 to 50 mg total daily dose, duloxetine 60 to 120 mg total daily dose, or venlafaxine 75 to 225 mg total daily dose) at a stable FDA approved dosage for at least the two consecutive months in the current episode immediately prior to the screening visit. Sertraline or citalopram are also permitted as background treatment for GAD at doses of 50 to 200 mg total daily dose and 20 to 40 mg total daily dose, respectively.

Exclusion criteria:

1. Subjects with a history of daily benzodiazepine use within one month of the screening visit.
2. Recent (defined as meeting disorder diagnostic criteria during the last 6 months) of a DSM IV TR Axis I diagnosis other than generalized anxiety disorder, with the following exceptions: a. Subjects with recent (in the last 2 months) major depressive disorder may be enrolled if the anxiety symptoms are predominant over the depressive symptoms, as judged by the Covi/Raskin criteria listed above and confirmed GAD as the primary diagnosis by the MINI structured interview. b. Comorbid social phobia and/or specific phobias are permitted as long as the anxiety symptoms due to these disorders are clinically less significant than the anxiety symptoms due to GAD and GAD is confirmed as the primary diagnosis by the MINI structured interview.
3. Recent (defined as meeting disorder diagnostic criteria during the last 6 months) of a DSM IV TR Axis I of panic disorder with or without agoraphobia, Post Traumatic Stress Disorder (PTSD), dissociative disorder, obsessive compulsive disorder, attention deficit disorder. If a subject has a past misdiagnosis of any of these disorders, or if the subject has another psychiatric disorder that in the opinion of the investigator affects the suitability of a subject for this study based on safety or other considerations, the investigator will need to contact the sponsor prior to screening.
4. Past and/or current DSM IV TR diagnosis of schizophrenia, schizoaffective disorder, other psychotic disorders, bipolar disorders (I or II), factitious disorder or cognitive disorder (including delirium, dementia, and amnestic disorder).
5. Presence of comorbid personality disorders (Axis II) based on DSM IV TR.
6. Subjects who meet DSM IV TR defined diagnostic criteria for psychoactive substance dependence (excluding nicotine dependence) within 12 months of screening or DSM IV TR defined substance abuse within 3 months prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (47):
- United States (47):
  - Comprehensive Clinical Development, Inc., Cerritos, California
  - Pharmacology Research Institute, Encino, California
  - Sun Valley Research Center, Imperial, California
  - Excell Research, Inc., Oceanside, California
  - NRC Research Institute, Orange, California
  - California Neuorpsychopharmacology Clinical Research Institute, LLC (CNRI-San Diego, LLC), San Diego, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Pacific Clinical Research Medical Group, Upland, California
  - Hartford Hospital, Hartford, Connecticut
  - Institute of Living, Hartford, Connecticut
  - Avail Clinical Research, LLC, DeLand, Florida
  - Gulfcoast Clinical Center, Fort Meyers, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Berma Research Group, Hialeah, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Sarkis Clinical Trials, Lake City, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Institute for Advanced Medical Research, Alpharetta, Georgia
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Northwest Behavioral Research Center, Roswell, Georgia
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Phoenix Medica Research, Inc, Prairie Village, Kansas
  - Pharmasite Research Inc, Baltimore, Maryland
  - Beacon Clinical Research, LLC, Brockton, Massachusetts
  - ActivMed Practices & Research, Inc, Methuen, Massachusetts
  - BCCR Trials, Natick, Massachusetts
  - Premier Psychiatric Research Institute. LLC., Lincoln, Nebraska
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Bio Behavioral Health, Toms River, New Jersey
  - SPRI Clinical Trials LLC, Brooklyn, New York
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - Comprehensive Clinical Development, Inc., Jamaica, New York
  - Bioscience Research LLC, Mount Kisco, New York
  - Fieve Clinical Research, Inc, New York, New York
  - Patient Priority Clinical Sites, LLC, Cincinnati, Ohio
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Summit Research Network (Oregon) Inc., Portland, Oregon
  - Suburban Research Associates, Media, Pennsylvania
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Futuresearch Trials of Dallas, Dallas, Texas
  - InSite Clinical Research, LLC, DeSoto, Texas
  - Family Psychiatry of The Woodlands, The Woodlands, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
  - Summit Research Network (Seattle) LLC, Seattle, Washington

REFERENCES:
- [Derived] Targum SD, Murphy C, Khan J, Zumpano L, Whitlock M, Simen AA, Binneman B. Audio Recording for Independent Confirmation of Clinical Assessments in Generalized Anxiety Disorder. Innov Clin Neurosci. 2018 Apr 1;15(3-4):37-42. PMID 29721364
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7431007&StudyName=An%208-week%2C%20Randomized%2C%20Phase%202%2C%20Double-blind%2C%20Sequential%20Parallel-group%20Comparison%20Study%20Of%20Two%20Dose%20Levels%20Of%20Pf%2006372865%20Compared%20To%20Placebo%20As%20An%20Adjunctive%20Treatment%20In%20Outpatients%20With%20Inadequate%20Response%20To%20Standard%20Of%20Care%20For%20Generalized%20Anxiety%20Disorder

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a sequential parallel study consisting of 2 stages: 4 week randomized treatment period (Stage 1) followed by a 4 week treatment period (Stage 2). Participants randomized to placebo for Stage 1, received either PF-06372865 or placebo in Stage 2 and participants randomized to PF-06372865 in Stage 1 were assigned to Placebo in Stage 2.
Groups:
- Placebo + Placebo: Participants received placebo matched to PF-06372865 twice daily for 4 weeks during Stage 1, followed by placebo matched to PF-06372865 twice daily for 4 weeks during Stage 2.
- Placebo + PF-06372865 2.5 mg: Participants received placebo matched to PF-06372865 twice daily for 4 weeks during Stage 1, followed by a single oral dose of PF-06372865 2.5 milligram (mg) tablet twice daily for 4 weeks during Stage 2.
- Placebo + PF-06372865 7.5 mg: Participants received placebo matched to PF-06372865 twice daily for 4 weeks during Stage 1, followed by single oral dose of PF-06372865 2.5 mg tablet twice daily for one week, then single oral dose of PF-06372865 7.5 mg tablet twice daily for 3 weeks during Stage 2.
- PF-06372865 2.5 mg + Placebo: Participants received single oral dose of PF-06372865 2.5 mg tablet twice daily for 4 weeks during Stage 1, followed by placebo matched to PF-06372865 twice daily for 4 weeks during Stage 2.
- PF-06372865 7.5 mg + Placebo: Participants received single oral dose of PF-06372865 2.5 mg tablet twice daily for one week, then PF-06372865 7.5 mg tablet twice daily for 3 weeks during Stage 1, followed by placebo matched to PF-06372865 twice daily for 4 weeks during Stage 2.
Period: Stage 1 ( 4 Weeks)
Arm/Group | Placebo + Placebo | Placebo + PF-06372865 2.5 mg | Placebo + PF-06372865 7.5 mg | PF-06372865 2.5 mg + Placebo | PF-06372865 7.5 mg + Placebo
Started | 15 | 15 | 15 | 24 | 21
Completed | 12 | 13 | 14 | 22 | 20
Not Completed | 3 | 2 | 1 | 2 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Participants | 1 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 1 | 0 | 0
Not completed — No Longer Meets Eligibility Criteria | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0
Period: Stage 2 (4 Weeks)
Arm/Group | Placebo + Placebo | Placebo + PF-06372865 2.5 mg | Placebo + PF-06372865 7.5 mg | PF-06372865 2.5 mg + Placebo | PF-06372865 7.5 mg + Placebo
Started | 12 | 13 | 14 | 22 | 20
Completed | 11 | 12 | 13 | 17 | 19
Not Completed | 1 | 1 | 1 | 5 | 1
Not completed — Withdrawal by Participants | 1 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 1 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo + PF-06372865 2.5 mg: Participants received placebo matched to PF-06372865 twice daily for 4 weeks during Stage 1, followed by a single oral dose of PF-06372865 2.5 mg tablet twice daily for 4 weeks during Stage 2.
- Total: Total of all reporting groups
Arm/Group | Placebo + Placebo | Placebo + PF-06372865 2.5 mg | Placebo + PF-06372865 7.5 mg | PF-06372865 2.5 mg + Placebo | PF-06372865 7.5 mg + Placebo | Total
Number analyzed (Participants) | 15 | 15 | 15 | 24 | 21 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (12.4) | 47.1 (15.6) | 42.7 (13.8) | 38.8 (14) | 42 (12) | 41.2 (13.7)
Gender [Count of Participants; unit: Participants]
  Female | 11 | 9 | 10 | 19 | 18 | 67
  Male | 4 | 6 | 5 | 5 | 3 | 23

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Anxiety Rating Scale (HAM-A) Total Scores at Baseline: Stage 1 and 2
Description: The HAM-A scale was a clinician rated interview scale designed to measure the signs and symptoms of anxiety. It had 14-items to rate the intensity of psychic and somatic anxiety on a 5-point severity scale. Each item ranging from 0 (not present) to 4 (very severe) were summed up to give a total possible score of 0 (not present) to 56 (very severe), where lower scores indicates less anxiety.
Time Frame: Stage 1: Baseline (Day 1 ), Stage 2: Baseline (Day 28)
Population: Stage 1 full analysis set: All randomized participants who received at least 1 dose of study treatment. Stage 2 placebo non-responder set: Subset of Stage 2 placebo set (participants who received placebo in Stage 1) with less than (<) 50% reduction in HAM-A during Stage 1 baseline,Week 4 and HAM-A value of greater than or equal to (>=)16 at Week 4.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo (Stage 1): All participants who received placebo matched to PF-06372865 2.5 mg or PF-06372865 7.5 mg, orally twice daily for 4 weeks during Stage 1.
- PF-06372865 2.5 mg (Stage 1): All participants who received a single dose of PF-06372865 2.5 mg tablet, orally twice daily for 4 weeks during Stage 1.
- PF-06372865 7.5 mg (Stage 1): All participants who received a single dose of PF-06372865 7.5 mg tablet, orally twice daily for 4 weeks during Stage 1.
- Placebo (Stage 2): All participants who received placebo matched to PF-06372865 2.5 mg or PF-06372865 7.5 mg, orally twice daily for 4 weeks during Stage 2.
- PF-06372865 2.5 mg (Stage 2): All participants who received a single dose of PF-06372865 2.5 mg tablet, twice daily for 4 weeks during Stage 2.
- PF-06372865 7.5 mg (Stage 2): All participants who received a single dose of PF-06372865 7.5 mg tablet, twice daily for 4 weeks during Stage 2.
Arm/Group | Placebo (Stage 1) | PF-06372865 2.5 mg (Stage 1) | PF-06372865 7.5 mg (Stage 1) | Placebo (Stage 2) | PF-06372865 2.5 mg (Stage 2) | PF-06372865 7.5 mg (Stage 2)
Number analyzed (Participants) | 45 | 24 | 21 | 6 | 8 | 8
units on a scale | 28 (4.48) | 26.7 (4.27) | 26.1 (4.0) | 26.2 (6.91) | 22.5 (4.24) | 22.5 (4.63)

2. Primary Outcome: Change From Baseline in Hamilton Anxiety Rating Scale (HAM-A) Total Scores at Week 4: Stage 1
Description: as for outcome 1
Time Frame: Week 4
Population: Full analysis set for Stage 1 included all randomized participants who had received at least 1 dose of randomized treatment. Here, number of participants analyzed (N) signifies those participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (Stage 1) | PF-06372865 2.5 mg (Stage 1) | PF-06372865 7.5 mg (Stage 1)
Number analyzed (Participants) | 40 | 22 | 20
units on a scale | -10.5 (1.16) | -7.9 (1.54) | -9.9 (1.62)
Statistical Analysis 1: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1); (PF-06372865 7.5 mg - Placebo). Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 1 was Day 1; Test type: Superiority or Other; p = 0.784, Mixed-Effects Model Repeated Measure; Least Square (LS) Mean Difference = 0.6, 90% CI 2-sided [-2.8 to 3.9], Standard Error of Mean 2.01
Statistical Analysis 2: Comparison: Placebo (Stage 1) vs PF-06372865 2.5 mg (Stage 1); (PF-06372865 2.5 mg - Placebo). Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 1 was Day 1; Test type: Superiority or Other; p = 0.184, Mixed-Effects Model Repeated Measure; LS Mean Difference = 2.6, 90% CI 2-sided [-0.6 to 5.8], Standard Error of Mean 1.94
Statistical Analysis 3: Comparison: PF-06372865 2.5 mg (Stage 1) vs PF-06372865 7.5 mg (Stage 1); (PF-06372865 7.5 mg - PF-06372865 2.5 mg). Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 1 was Day 1; Test type: Superiority or Other; p = 0.360, Mixed-Effects Model Repeated Measure; LS Mean Difference = -2.0, 90% CI 2-sided [-5.7 to 1.6], Standard Error of Mean 2.22

3. Primary Outcome: Hamilton Anxiety Rating Scale (HAM-A) Total Scores at Week 4 During Stage 1 and at Week 8 During Stage 2
Description: as for outcome 1
Time Frame: Stage 1: Week 4, Stage 2: Week 8
Population: Full analysis set for Stage 1 and Placebo Non-Responder set for Stage 2. Here, 'N' signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Stage 1) | PF-06372865 2.5 mg (Stage 1) | PF-06372865 7.5 mg (Stage 1) | Placebo (Stage 2) | PF-06372865 2.5 mg (Stage 2) | PF-06372865 7.5 mg (Stage 2)
Number analyzed (Participants) | 40 | 22 | 20 | 6 | 8 | 7
units on a scale | 17.5 (8.03) | 18.7 (9.49) | 16.5 (6.87) | 21.7 (9.44) | 15.5 (7.01) | 19.4 (8.44)

4. Secondary Outcome: Change From Baseline in Hamilton Anxiety Rating Scale (HAM-A) Total Scores at Week 5, Week 6, Week 7 and Week 8: Stage 2
Description: as for outcome 1
Time Frame: Week 5, 6, 7, 8
Population: Stage 2 placebo non-responder set: Subset of Stage 2 placebo set (participants who received placebo in Stage 1) < 50 % reduction in HAM-A during Stage 1 baseline, Week 4 and HAM-A value of >=16 at Week 4. Here, 'n' signifies those participants who were evaluable at specified time point for each arm, respectively.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (Stage 2) | PF-06372865 2.5 mg (Stage 2) | PF-06372865 7.5 mg (Stage 2)
Number analyzed (Participants) | 6 | 8 | 8
units on a scale
  Week 5 (n = 6, 8, 8) | -0.4 (1.77) | -1.5 (1.49) | 0.5 (1.49)
  Week 6 (n = 6, 8, 8) | -3.3 (2.25) | -0.8 (1.89) | -1.2 (1.89)
  Week 7 (n = 6, 8, 7) | -4.6 (2.02) | -4.4 (1.70) | -1.9 (1.74)
  Week 8 (n = 6, 8, 7) | -4.1 (2.92) | -7.2 (2.46) | -3.4 (2.54)
Statistical Analysis 1: Comparison: Placebo (Stage 2) vs PF-06372865 7.5 mg (Stage 2); (PF-06372865 7.5 mg - Placebo). Week 5: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 2 was Week 4 (Day 28); Test type: Superiority or Other; p = 0.708, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.9, 90% CI 2-sided [-3.2 to 5.0], Standard Error of Mean 2.36
Statistical Analysis 2: Comparison: Placebo (Stage 2) vs PF-06372865 2.5 mg (Stage 2); (PF-06372865 2.5 mg - Placebo). Week 5: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 2 was Week 4 (Day 28); Test type: Superiority or Other; p = 0.646, Mixed-Effects Model Repeated Measure; LS Mean Difference = -1.1, 90% CI 2-sided [-5.2 to 3.0], Standard Error of Mean 2.36
Statistical Analysis 3: Comparison: PF-06372865 2.5 mg (Stage 2) vs PF-06372865 7.5 mg (Stage 2); (PF-06372865 7.5 mg - PF-06372865 2.5 mg). Week 5: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 2 was Week 4 (Day 28); Test type: Superiority or Other; p = 0.352, Mixed-Effects Model Repeated Measure; LS Mean Difference = 2.0, 90% CI 2-sided [-1.6 to 5.6], Standard Error of Mean 2.09
Statistical Analysis 4: Comparison: Placebo (Stage 2) vs PF-06372865 7.5 mg (Stage 2); (PF-06372865 7.5 mg - Placebo). Week 6: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 2 was Week 4 (Day 28); Test type: Superiority or Other; p = 0.495, Mixed-Effects Model Repeated Measure; LS Mean Difference = 2.1, 90% CI 2-sided [-3.1 to 7.3], Standard Error of Mean 2.99
Statistical Analysis 5: Comparison: Placebo (Stage 2) vs PF-06372865 2.5 mg (Stage 2); (PF-06372865 2.5 mg - Placebo). Week 6: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 2 was Week 4 (Day 28); Test type: Superiority or Other; p = 0.422, Mixed-Effects Model Repeated Measure; LS Mean Difference = 2.5, 90% CI 2-sided [-2.7 to 7.6], Standard Error of Mean 2.99
Statistical Analysis 6: Comparison: PF-06372865 2.5 mg (Stage 2) vs PF-06372865 7.5 mg (Stage 2); (PF-06372865 7.5 mg - PF-06372865 2.5 mg). Week 6: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 2 was Week 4 (Day 28); Test type: Superiority or Other; p = 0.889, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.4, 90% CI 2-sided [-5.0 to 4.2], Standard Error of Mean 2.65
Statistical Analysis 7: Comparison: Placebo (Stage 2) vs PF-06372865 7.5 mg (Stage 2); (PF-06372865 7.5 mg - Placebo). Week 7: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 2 was Week 4 (Day 28); Test type: Superiority or Other; p = 0.324, Mixed-Effects Model Repeated Measure; LS Mean Difference = 2.7, 90% CI [-2.0 to 7.4], Standard Error of Mean 2.71
Statistical Analysis 8: Comparison: Placebo (Stage 2) vs PF-06372865 2.5 mg (Stage 2); (PF-06372865 2.5 mg - Placebo). Week 7: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 2 was Week 4 (Day 28); Test type: Superiority or Other; p = 0.939, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.2, 90% CI 2-sided [-4.5 to 4.9], Standard Error of Mean 2.69
Statistical Analysis 9: Comparison: PF-06372865 2.5 mg (Stage 2) vs PF-06372865 7.5 mg (Stage 2); (PF-06372865 7.5 mg - PF-06372865 2.5 mg). Week 7: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 2 was Week 4 (Day 28); Test type: Superiority or Other; p = 0.308, Mixed-Effects Model Repeated Measure; LS Mean Difference = 2.5, 90% CI 2-sided [-1.7 to 6.7], Standard Error of Mean 2.42
Statistical Analysis 10: Comparison: Placebo (Stage 2) vs PF-06372865 7.5 mg (Stage 2); (PF-06372865 7.5 mg - Placebo). Week 8: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 2 was Week 4 (Day 28); Test type: Superiority or Other; p = 0.846, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.8, 90% CI 2-sided [-6.0 to 7.6], Standard Error of Mean 3.92
Statistical Analysis 11: Comparison: Placebo (Stage 2) vs PF-06372865 2.5 mg (Stage 2); (PF-06372865 2.5 mg - Placebo). Week 8: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 2 was Week 4 (Day 28); Test type: Superiority or Other; p = 0.449, Mixed-Effects Model Repeated Measure; LS Mean Difference = -3.0, 90% CI 2-sided [-9.8 to 3.7], Standard Error of Mean 3.89
Statistical Analysis 12: Comparison: PF-06372865 2.5 mg (Stage 2) vs PF-06372865 7.5 mg (Stage 2); (PF-06372865 7.5 mg - PF-06372865 2.5 mg). Week 8: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 2 was Week 4 (Day 28); Test type: Superiority or Other; p = 0.295, Mixed-Effects Model Repeated Measure; LS Mean Difference = 3.8, 90% CI 2-sided [-2.3 to 9.9], Standard Error of Mean 3.51

5. Secondary Outcome: Sheehan Disability Scale (SDS) Total Score and Social, Work, Family Subscale Scores at Baseline: Stage 1 and Stage 2
Description: SDS was a copyrighted, three question instrument designed to assess functional impairment associated with mental disorders in three domains: work impairment, social impairment, and impairment of family life or home responsibilities. Disability scores were reported for each of the questions (subscale scores range from 0 to 10) and a total disability score was calculated as the sum of scores for each question (total scores range from 0 to 30). Higher scores reflect greater impairment.
Time Frame: Stage 1: Baseline (Day 1 ), Stage 2: Baseline (Day 28)
Population: Full analysis set for Stage 1 and Placebo Non-Responder set for Stage 2. Here, 'n' signifies those participants who were evaluable at specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Stage 1) | PF-06372865 2.5 mg (Stage 1) | PF-06372865 7.5 mg (Stage 1) | Placebo (Stage 2) | PF-06372865 2.5 mg (Stage 2) | PF-06372865 7.5 mg (Stage 2)
Number analyzed (Participants) | 45 | 24 | 21 | 6 | 8 | 8
units on a scale
  Total Score (n=45,24,21,6,8,8) | 18.6 (5.80) | 19.6 (5.73) | 17.0 (5.55) | 23.0 (2.76) | 15.3 (6.86) | 17.4 (4.89)
  Social Subscale Score (n=45,24,21,6,8,8) | 6.6 (1.96) | 7.2 (1.88) | 5.9 (1.80) | 7.8 (1.17) | 5.0 (2.56) | 5.5 (1.20)
  Work Subscale Score (n =37,19,16,6,6,7) | 5.9 (2.59) | 5.8 (3.06) | 5.9 (2.28) | 7.5 (1.38) | 5.3 (2.58) | 5.6 (2.44)
  Family Subscale Score (n= 45,24,21,6,8,8) | 6.2 (2.10) | 6.2 (2.17) | 5.5 (2.23) | 7.7 (1.03) | 5.3 (2.49) | 6.3 (2.60)

6. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Total Score and Social, Work, Family Subscale Scores: Stage 1 and Stage 2
Description: as for outcome 5
Time Frame: Stage 1: Week 4, Stage 2: Week 8
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (Stage 1) | PF-06372865 2.5 mg (Stage 1) | PF-06372865 7.5 mg (Stage 1) | Placebo (Stage 2) | PF-06372865 2.5 mg (Stage 2) | PF-06372865 7.5 mg (Stage 2)
Number analyzed (Participants) | 45 | 24 | 21 | 6 | 8 | 8
units on a scale
  Total Score (n= 40,22,20,6,8,7) | -3.5 (0.98) | -5.3 (1.33) | -4.7 (1.40) | -3.5 (2.90) | -5.9 (2.36) | -2.4 (2.40)
  Social Sub-scale Score (n= 40,22,20,6,8,7) | -1.8 (0.53) | -1.7 (0.50) | -1.8 (0.53) | -0.3 (1.32) | -2.3 (1.03) | -0.6 (1.07)
  Work Sub-scale Score (n= 30,16,14,6,5,6) | -0.7 (0.41) | -2.4 (0.56) | -1.5 (0.60) | -0.7 (0.96) | -2.6 (1.01) | -1.4 (0.93)
  Family Sub-scale Score 9 (n= 40, 22, 20,6,8,7) | -0.9 (0.36) | -1.6 (0.48) | -1.4 (0.51) | -1.4 (0.92) | -1.9 (0.78) | -1.0 (0.80)
Statistical Analysis 1: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1); (PF-06372865 7.5 mg - Placebo). Total Score (Week 4): The ANCOVA model included change from baseline as dependent variable, and treatment and baseline in the model. Baseline for Stage 1 is Day 1 and baseline for Stage 2 is Week 4 (Day 28). The estimates from Stage 1 and the Stage 2 were combined together using a weighted mean (weight=0.5) and assuming the covariance between the two treatment effect estimates is zero; Test type: Superiority or Other; p = 0.514, ANCOVA; Least Squares Mean Difference = -1.1, 90% CI 2-sided [-4.0 to 1.7], Standard Error of Mean 1.72
Statistical Analysis 2: Comparison: Placebo (Stage 1) vs PF-06372865 2.5 mg (Stage 1); (PF-06372865 2.5 mg - Placebo). Total Score (Week 4): The ANCOVA model included change from baseline as dependent variable, and treatment and baseline in the model. Baseline for Stage 1 is Day 1 and baseline for Stage 2 is Week 4 (Day 28). The estimates from Stage 1 and the Stage 2 were combined together using a weighted mean (weight=0.5) and assuming the covariance between the two treatment effect estimates is zero; Test type: Superiority or Other; p = 0.302, ANCOVA; LS Mean Difference = -1.7, 90% CI 2-sided [-4.5 to 1.0], Standard Error of Mean 1.65
Statistical Analysis 3: Comparison: PF-06372865 2.5 mg (Stage 1) vs PF-06372865 7.5 mg (Stage 1); (PF-06372865 7.5 mg - PF-06372865 2.5 mg). Total Score (Week 4): The ANCOVA model included change from baseline as dependent variable, and treatment and baseline in the model. Baseline for Stage 1 is Day 1 and baseline for Stage 2 is Week 4 (Day 28). The estimates from Stage 1 and the Stage 2 were combined together using a weighted mean (weight=0.5) and assuming the covariance between the two treatment effect estimates is zero; Test type: Superiority or Other; p = 0.736, ANCOVA; LS Mean Difference = 0.6, 90% CI 2-sided [-2.6 to 3.8], Standard Error of Mean 1.94
Statistical Analysis 4: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1); (PF-06372865 7.5 mg - Placebo). Total Score (Week 8): The ANCOVA model included change from baseline as dependent variable, and treatment and baseline in the model. Baseline for Stage 1 is Day 1 and baseline for Stage 2 is Week 4 (Day 28). The estimates from Stage 1 and the Stage 2 were combined together using a weighted mean (weight=0.5) and assuming the covariance between the two treatment effect estimates is zero; Test type: Superiority or Other; p = 0.775, ANCOVA; LS Mean Difference = 1.1, 90% CI 2-sided [-5.6 to 7.8], Standard Error of Mean 3.85
Statistical Analysis 5: Comparison: Placebo (Stage 1) vs PF-06372865 2.5 mg (Stage 1); (PF-06372865 2.5 mg - Placebo). Total Score (Week 8): The ANCOVA model included change from baseline as dependent variable, and treatment and baseline in the model. Baseline for Stage 1 is Day 1 and baseline for Stage 2 is Week 4 (Day 28). The estimates from Stage 1 and the Stage 2 were combined together using a weighted mean (weight=0.5) and assuming the covariance between the two treatment effect estimates is zero; Test type: Superiority or Other; p = 0.553, ANCOVA; LS Mean Difference = -2.4, 90% CI 2-sided [-9.4 to 4.5], Standard Error of Mean 4.00
Statistical Analysis 6: Comparison: PF-06372865 2.5 mg (Stage 1) vs PF-06372865 7.5 mg (Stage 1); (PF-06372865 7.5 mg - PF-06372865 2.5 mg). Total Score ( Week 8): The ANCOVA model included change from baseline as dependent variable, and treatment and baseline in the model. Baseline for Stage 1 is Day 1 and baseline for Stage 2 is Week 4 (Day 28). The estimates from Stage 1 and the Stage 2 were combined together using a weighted mean (weight=0.5) and assuming the covariance between the two treatment effect estimates is zero; Test type: Superiority or Other; p = 0.299, ANCOVA; LS Mean Difference = 3.5, 90% CI 2-sided [-2.2 to 9.3], Standard Error of Mean 3.30
Statistical Analysis 7: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1); (PF-06372865 7.5 mg - Placebo). Social Sub-Scale Score (Week 4): The ANCOVA model included change from baseline as dependent variable, and treatment and baseline in the model. Baseline for Stage 1 is Day 1 and baseline for Stage 2 is Week 4 (Day 28). The estimates from Stage 1 and the Stage 2 were combined together using a weighted mean (weight=0.5) and assuming the covariance between the two treatment effect estimates is zero; Test type: Superiority or Other; p = 0.994, ANCOVA; LS Mean Difference = 0.0, 90% CI 2-sided [-1.1 to 1.1], Standard Error of Mean 0.65
Statistical Analysis 8: Comparison: Placebo (Stage 1) vs PF-06372865 2.5 mg (Stage 1); (PF-06372865 2.5 mg - Placebo). Social Sub-Scale Score (Week 4): The ANCOVA model included change from baseline as dependent variable, and treatment and baseline in the model. Baseline for Stage 1 is Day 1 and baseline for Stage 2 is Week 4 (Day 28). The estimates from Stage 1 and the Stage 2 were combined together using a weighted mean (weight=0.5) and assuming the covariance between the two treatment effect estimates is zero; Test type: Superiority or Other; p = 0.870, ANCOVA; LS Mean Difference = 0.1, 90% CI 2-sided [-0.9 to 1.1], Standard Error of Mean 0.62
Statistical Analysis 9: Comparison: PF-06372865 2.5 mg (Stage 1) vs PF-06372865 7.5 mg (Stage 1); (PF-06372865 7.5 mg - PF-06372865 2.5 mg). Social Sub-Scale Score (Week 4): The ANCOVA model included change from baseline as dependent variable, and treatment and baseline in the model. Baseline for Stage 1 is Day 1 and baseline for Stage 2 is Week 4 (Day 28). The estimates from Stage 1 and the Stage 2 were combined together using a weighted mean (weight=0.5) and assuming the covariance between the two treatment effect estimates is zero; Test type: Superiority or Other; p = 0.885, ANCOVA; LS Mean Difference = -0.1, 90% CI 2-sided [-1.3 to 1.1], Standard Error of Mean 0.74
Statistical Analysis 10: Comparison: Placebo (Stage 2) vs PF-06372865 7.5 mg (Stage 2); (PF-06372865 7.5 mg - Placebo). Social Sub-Scale Score (Week 8): The ANCOVA model included change from baseline as dependent variable, and treatment and baseline in the model. Baseline for Stage 1 is Day 1 and baseline for Stage 2 is Week 4 (Day 28). The estimates from Stage 1 and the Stage 2 were combined together using a weighted mean (weight=0.5) and assuming the covariance between the two treatment effect estimates is zero; Test type: Superiority or Other; p = 0.834, ANCOVA; LS Mean Difference = -0.4, 90% CI 2-sided [-3.5 to 2.7], Standard Error of Mean 1.78
Statistical Analysis 11: Comparison: Placebo (Stage 2) vs PF-06372865 2.5 mg (Stage 2); (PF-06372865 2.5 mg - Placebo). Social Sub-Scale Score (Week 8): The ANCOVA model included change from baseline as dependent variable, and treatment and baseline in the model. Baseline for Stage 1 is Day 1 and baseline for Stage 2 is Week 4 (Day 28). The estimates from Stage 1 and the Stage 2 were combined together using a weighted mean (weight=0.5) and assuming the covariance between the two treatment effect estimates is zero; Test type: Superiority or Other; p = 0.281, ANCOVA; LS Mean Difference = -2.0, 90% CI 2-sided [-5.1 to 1.1], Standard Error of Mean 1.80
Statistical Analysis 12: Comparison: PF-06372865 2.5 mg (Stage 2) vs PF-06372865 7.5 mg (Stage 2); (PF-06372865 7.5 mg - PF-06372865 2.5 mg). Social Sub-Scale Score (Week 8): The ANCOVA model included change from baseline as dependent variable, and treatment and baseline in the model. Baseline for Stage 1 is Day 1 and baseline for Stage 2 is Week 4 (Day 28). The estimates from Stage 1 and the Stage 2 were combined together using a weighted mean (weight=0.5) and assuming the covariance between the two treatment effect estimates is zero; Test type: Superiority or Other; p = 0.272, ANCOVA; LS Mean Difference = 1.6, 90% CI 2-sided [-0.9 to 4.1], Standard Error of Mean 1.43
Statistical Analysis 13: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1); (PF-06372865 7.5 mg - Placebo). Work Sub-Scale Score (Week 4): The ANCOVA model included change from baseline as dependent variable, and treatment and baseline in the model. Baseline for Stage 1 is Day 1 and baseline for Stage 2 is Week 4 (Day 28). The estimates from Stage 1 and the Stage 2 were combined together using a weighted mean (weight=0.5) and assuming the covariance between the two treatment effect estimates is zero; Test type: Superiority or Other; p = 0.249, ANCOVA; LS Mean Difference = -0.8, 90% CI 2-sided [-2.1 to 0.4], Standard Error of Mean 0.73
Statistical Analysis 14: Comparison: Placebo (Stage 1) vs PF-06372865 2.5 mg (Stage 1); (PF-06372865 2.5 mg - Placebo). Work Sub-Scale Score (Week 4): The ANCOVA model included change from baseline as dependent variable, and treatment and baseline in the model. Baseline for Stage 1 is Day 1 and baseline for Stage 2 is Week 4 (Day 28). The estimates from Stage 1 and the Stage 2 were combined together using a weighted mean (weight=0.5) and assuming the covariance between the two treatment effect estimates is zero; Test type: Superiority or Other; p = 0.016, ANCOVA; LS Mean Difference = -1.7, 90% CI 2-sided [-2.9 to -0.6], Standard Error of Mean 0.70
Statistical Analysis 15: Comparison: PF-06372865 2.5 mg (Stage 1) vs PF-06372865 7.5 mg (Stage 1); (PF-06372865 7.5 mg - PF-06372865 2.5 mg). Work Sub-Scale Score (Week 4): The ANCOVA model included change from baseline as dependent variable, and treatment and baseline in the model. Baseline for Stage 1 is Day 1 and baseline for Stage 2 is Week 4 (Day 28). The estimates from Stage 1 and the Stage 2 were combined together using a weighted mean (weight=0.5) and assuming the covariance between the two treatment effect estimates is zero; Test type: Superiority or Other; p = 0.285, ANCOVA; LS Mean Difference = 0.9, 0.285% CI 2-sided [-0.5 to 2.3], Standard Error of Mean 0.82
Statistical Analysis 16: Comparison: Placebo (Stage 2) vs PF-06372865 7.5 mg (Stage 2); (PF-06372865 7.5 mg - Placebo). Work Sub-Scale Score ( Week 8): The ANCOVA model included change from baseline as dependent variable, and treatment and baseline in the model. Baseline for Stage 1 is Day 1 and baseline for Stage 2 is Week 4 (Day 28). The estimates from Stage 1 and the Stage 2 were combined together using a weighted mean (weight=0.5) and assuming the covariance between the two treatment effect estimates is zero; Test type: Superiority or Other; p = 0.635, ANCOVA; LS Mean Difference = -0.7, 90% CI 2-sided [-3.1 to 1.8], Standard Error of Mean 1.38
Statistical Analysis 17: Comparison: Placebo (Stage 2) vs PF-06372865 2.5 mg (Stage 2); (PF-06372865 2.5 mg - Placebo). Work Sub-Scale Score (Week 8): The ANCOVA model included change from baseline as dependent variable, and treatment and baseline in the model. Baseline for Stage 1 is Day 1 and baseline for Stage 2 is Week 4 (Day 28). The estimates from Stage 1 and the Stage 2 were combined together using a weighted mean (weight=0.5) and assuming the covariance between the two treatment effect estimates is zero; Test type: Superiority or Other; p = 0.217, ANCOVA; LS Mean Difference = -1.9, 90% CI 2-sided [-4.4 to 0.7], Standard Error of Mean 1.43
Statistical Analysis 18: Comparison: PF-06372865 2.5 mg (Stage 2) vs PF-06372865 7.5 mg (Stage 2); (PF-06372865 7.5 mg - PF-06372865 2.5 mg). Work Sub-Scale Score (Week 8): The ANCOVA model included change from baseline as dependent variable, and treatment and baseline in the model. Baseline for Stage 1 is Day 1 and baseline for Stage 2 is Week 4 (Day 28). The estimates from Stage 1 and the Stage 2 were combined together using a weighted mean (weight=0.5) and assuming the covariance between the two treatment effect estimates is zero; Test type: Superiority or Other; p = 0.399, ANCOVA; LS Mean Difference = 1.2, 90% CI 2-sided [-1.2 to 3.6], Standard Error of Mean 1.36
Statistical Analysis 19: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1); (PF-06372865 7.5 mg - Placebo). Family Sub-Scale Score (Week 4): The ANCOVA model included change from baseline as dependent variable, and treatment and baseline in the model. Baseline for Stage 1 is Day 1 and baseline for Stage 2 is Week 4 (Day 28). The estimates from Stage 1 and the Stage 2 were combined together using a weighted mean (weight=0.5) and assuming the covariance between the two treatment effect estimates is zero; Test type: Superiority or Other; p = 0.429, ANCOVA; LS Mean Difference = -0.5, 90% CI 2-sided [-1.5 to 0.5], Standard Error of Mean 0.62
Statistical Analysis 20: Comparison: Placebo (Stage 1) vs PF-06372865 2.5 mg (Stage 1); (PF-06372865 2.5 mg - Placebo). Family Sub-Scale Score (Week 4): The ANCOVA model included change from baseline as dependent variable, and treatment and baseline in the model. Baseline for Stage 1 is Day 1 and baseline for Stage 2 is Week 4 (Day 28). The estimates from Stage 1 and the Stage 2 were combined together using a weighted mean (weight=0.5) and assuming the covariance between the two treatment effect estimates is zero; Test type: Superiority or Other; p = 0.260, ANCOVA; LS Mean Difference = -0.7, 90% CI 2-sided [-1.7 to 0.3], Standard Error of Mean 0.60
Statistical Analysis 21: Comparison: PF-06372865 2.5 mg (Stage 1) vs PF-06372865 7.5 mg (Stage 1); (PF-06372865 7.5 mg - PF-06372865 2.5 mg). Family Sub-Scale Score (Week 4): The ANCOVA model included change from baseline as dependent variable, and treatment and baseline in the model. Baseline for Stage 1 is Day 1 and baseline for Stage 2 is Week 4 (Day 28). The estimates from Stage 1 and the Stage 2 were combined together using a weighted mean (weight=0.5) and assuming the covariance between the two treatment effect estimates is zero; Test type: Superiority or Other; p = 0.799, ANCOVA; LS Mean Difference = 0.2, 90% CI 2-sided [-1.0 to 1.3], Standard Error of Mean 0.70
Statistical Analysis 22: Comparison: Placebo (Stage 2) vs PF-06372865 7.5 mg (Stage 2); (PF-06372865 7.5 mg - Placebo). Family Sub-Scale Score (Week 8): The ANCOVA model included change from baseline as dependent variable, and treatment and baseline in the model. Baseline for Stage 1 is Day 1 and baseline for Stage 2 is Week 4 (Day 28). The estimates from Stage 1 and the Stage 2 were combined together using a weighted mean (weight=0.5) and assuming the covariance between the two treatment effect estimates is zero; Test type: Superiority or Other; p = 0.738, ANCOVA; LS Mean Difference = 0.4, 90% CI 2-sided [-1.7 to 2.5], Standard Error of Mean 1.22
Statistical Analysis 23: Comparison: Placebo (Stage 2) vs PF-06372865 2.5 mg (Stage 2); (PF-06372865 2.5 mg - Placebo). Family Sub-Scale Score (Week 8): The ANCOVA model included change from baseline as dependent variable, and treatment and baseline in the model. Baseline for Stage 1 is Day 1 and baseline for Stage 2 is Week 4 (Day 28). The estimates from Stage 1 and the Stage 2 were combined together using a weighted mean (weight=0.5) and assuming the covariance between the two treatment effect estimates is zero; Test type: Superiority or Other; p = 0.691, ANCOVA; LS Mean Difference = 1.26, 90% CI 2-sided [-2.7 to 1.7], Standard Error of Mean -0.5
Statistical Analysis 24: Comparison: PF-06372865 2.5 mg (Stage 2) vs PF-06372865 7.5 mg (Stage 2); (PF-06372865 7.5 mg - PF-06372865 2.5 mg). Family Sub-Scale Score (Week 8): The ANCOVA model included change from baseline as dependent variable, and treatment and baseline in the model. Baseline for Stage 1 is Day 1 and baseline for Stage 2 is Week 4 (Day 28). The estimates from Stage 1 and the Stage 2 were combined together using a weighted mean (weight=0.5) and assuming the covariance between the two treatment effect estimates is zero; Test type: Superiority or Other; p = 0.417, ANCOVA; LS Mean Difference = 0.9, 90% CI 2-sided [-1.0 to 2.9], Standard Error of Mean 1.11
Statistical Analysis 25: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1) vs Placebo (Stage 2) vs PF-06372865 7.5 mg (Stage 2); (PF-06372865 7.5 mg - Placebo). Total Score (Combined Stage 1 and Stage 2): The ANCOVA model included change from baseline as dependent variable, and treatment and baseline in the model. Baseline for Stage 1 is Day 1 and baseline for Stage 2 is Week 4 (Day 28). The estimates from Stage 1 and the Stage 2 were combined together using a weighted mean (weight=0.5) and assuming the covariance between the two treatment effect estimates is zero; Test type: Superiority or Other; p = 0.998, ANCOVA; LS Mean Difference = 0.0, 90% CI 2-sided [-3.7 to 3.7], Standard Error of Mean 2.11
Statistical Analysis 26: Comparison: Placebo (Stage 1) vs PF-06372865 2.5 mg (Stage 1) vs Placebo (Stage 2) vs PF-06372865 2.5 mg (Stage 2); (PF-06372865 2.5 mg - Placebo). Total Score (Combined Stage 1 and Stage 2): The ANCOVA model included change from baseline as dependent variable, and treatment and baseline in the model. Baseline for Stage 1 is Day 1 and baseline for Stage 2 is Week 4 (Day 28). The estimates from Stage 1 and the Stage 2 were combined together using a weighted mean (weight=0.5) and assuming the covariance between the two treatment effect estimates is zero; Test type: Superiority or Other; p = 0.353, ANCOVA; LS Mean Difference = -2.1, 90% CI 2-sided [-5.8 to 1.7], Standard Error of Mean 2.16
Statistical Analysis 27: Comparison: PF-06372865 2.5 mg (Stage 1) vs PF-06372865 7.5 mg (Stage 1) vs PF-06372865 2.5 mg (Stage 2) vs PF-06372865 7.5 mg (Stage 2); (PF-06372865 7.5 mg - PF-06372865 2.5 mg). Total Score (Combined Stage 1 and Stage 2): The ANCOVA model included change from baseline as dependent variable, and treatment and baseline in the model. Baseline for Stage 1 is Day 1 and baseline for Stage 2 is Week 4 (Day 28). The estimates from Stage 1 and the Stage 2 were combined together using a weighted mean (weight=0.5) and assuming the covariance between the two treatment effect estimates is zero; Test type: Superiority or Other; p = 0.296, ANCOVA; LS Mean Difference = 2.1, 90% CI 2-sided [-1.3 to 5.4], Standard Error of Mean 1.92
Statistical Analysis 28: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1) vs Placebo (Stage 2) vs PF-06372865 7.5 mg (Stage 2); (PF-06372865 7.5 mg - Placebo). Social Sub-Scale Score (Combined Stage 1 and Stage 2): The ANCOVA model included change from baseline as dependent variable, and treatment and baseline in the model. Baseline for Stage 1 is Day 1 and baseline for Stage 2 is Week 4 (Day 28). The estimates from Stage 1 and the Stage 2 were combined together using a weighted mean (weight=0.5) and assuming the covariance between the two treatment effect estimates is zero; Test type: Superiority or Other; p = 0.841, ANCOVA; LS Mean Difference = -0.2, 90% CI 2-sided [-1.8 to 1.5], Standard Error of Mean 0.95
Statistical Analysis 29: Comparison: Placebo (Stage 1) vs PF-06372865 2.5 mg (Stage 1) vs Placebo (Stage 2) vs PF-06372865 2.5 mg (Stage 2); (PF-06372865 2.5 mg - Placebo). Social Sub-Scale Score (Combined Stage 1 and Stage 2): The ANCOVA model included change from baseline as dependent variable, and treatment and baseline in the model. Baseline for Stage 1 is Day 1 and baseline for Stage 2 is Week 4 (Day 28). The estimates from Stage 1 and the Stage 2 were combined together using a weighted mean (weight=0.5) and assuming the covariance between the two treatment effect estimates is zero; Test type: Superiority or Other; p = 0.332, ANCOVA; LS Mean Difference = -1.0, 90% CI 2-sided [-2.6 to 0.7], Standard Error of Mean 0.95
Statistical Analysis 30: Comparison: PF-06372865 2.5 mg (Stage 1) vs PF-06372865 7.5 mg (Stage 1) vs PF-06372865 2.5 mg (Stage 2) vs PF-06372865 7.5 mg (Stage 2); (PF-06372865 7.5 mg - PF-06372865 2.5 mg). Social Sub-Scale Score (Combined Stage 1 and Stage 2): The ANCOVA model included change from baseline as dependent variable, and treatment and baseline in the model. Baseline for Stage 1 is Day 1 and baseline for Stage 2 is Week 4 (Day 28). The estimates from Stage 1 and the Stage 2 were combined together using a weighted mean (weight=0.5) and assuming the covariance between the two treatment effect estimates is zero; Test type: Superiority or Other; p = 0.359, ANCOVA; LS Mean Difference = 0.8, 90% CI 2-sided [-0.6 to 2.2], Standard Error of Mean 0.81
Statistical Analysis 31: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1) vs Placebo (Stage 2) vs PF-06372865 7.5 mg (Stage 2); (PF-06372865 7.5 mg - Placebo). Work Sub-Scale Score (Combined Stage 1 and Stage 2): The ANCOVA model included change from baseline as dependent variable, and treatment and baseline in the model. Baseline for Stage 1 is Day 1 and baseline for Stage 2 is Week 4 (Day 28). The estimates from Stage 1 and the Stage 2 were combined together using a weighted mean (weight=0.5) and assuming the covariance between the two treatment effect estimates is zero; Test type: Superiority or Other; p = 0.347, ANCOVA; LS Mean Difference = -0.8, 90% CI 2-sided [-2.1 to 0.6], Standard Error of Mean 0.78
Statistical Analysis 32: Comparison: Placebo (Stage 1) vs PF-06372865 2.5 mg (Stage 1) vs Placebo (Stage 2) vs PF-06372865 2.5 mg (Stage 2); (PF-06372865 2.5 mg - Placebo). Work Sub-Scale Score (Combined Stage 1 and Stage 2): The ANCOVA model included change from baseline as dependent variable, and treatment and baseline in the model. Baseline for Stage 1 is Day 1 and baseline for Stage 2 is Week 4 (Day 28). The estimates from Stage 1 and the Stage 2 were combined together using a weighted mean (weight=0.5) and assuming the covariance between the two treatment effect estimates is zero; Test type: Superiority or Other; p = 0.041, ANCOVA; LS Mean Difference = -1.8, 90% CI 2-sided [-3.2 to -0.4], Standard Error of Mean 0.80
Statistical Analysis 33: Comparison: PF-06372865 2.5 mg (Stage 1) vs PF-06372865 7.5 mg (Stage 1) vs PF-06372865 2.5 mg (Stage 2) vs PF-06372865 7.5 mg (Stage 2); (PF-06372865 7.5 mg - PF-06372865 2.5 mg). Work Sub-Scale Score (Combined Stage 1 and Stage 2): The ANCOVA model included change from baseline as dependent variable, and treatment and baseline in the model. Baseline for Stage 1 is Day 1 and baseline for Stage 2 is Week 4 (Day 28). The estimates from Stage 1 and the Stage 2 were combined together using a weighted mean (weight=0.5) and assuming the covariance between the two treatment effect estimates is zero; Test type: Superiority or Other; p = 0.212, ANCOVA; LS Mean Difference = 1.0, 90% CI 2-sided [-0.4 to 2.4], Standard Error of Mean 0.79
Statistical Analysis 34: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1) vs Placebo (Stage 2) vs PF-06372865 7.5 mg (Stage 2); (PF-06372865 7.5 mg - Placebo). Family Sub-Scale Score (Combined Stage 1 and Stage 2): The ANCOVA model included change from baseline as dependent variable, and treatment and baseline in the model. Baseline for Stage 1 is Day 1 and baseline for Stage 2 is Week 4 (Day 28). The estimates from Stage 1 and the Stage 2 were combined together using a weighted mean (weight=0.5) and assuming the covariance between the two treatment effect estimates is zero; Test type: Superiority or Other; p = 0.954, ANCOVA; LS Mean Difference = 0.0, 90% CI 2-sided [-1.2 to 1.2], Standard Error of Mean 0.69
Statistical Analysis 35: Comparison: Placebo (Stage 1) vs PF-06372865 2.5 mg (Stage 1) vs Placebo (Stage 2) vs PF-06372865 2.5 mg (Stage 2); (PF-06372865 2.5 mg - Placebo). Family Sub-Scale Score (Combined Stage 1 and Stage 2): The ANCOVA model included change from baseline as dependent variable, and treatment and baseline in the model. Baseline for Stage 1 is Day 1 and baseline for Stage 2 is Week 4 (Day 28). The estimates from Stage 1 and the Stage 2 were combined together using a weighted mean (weight=0.5) and assuming the covariance between the two treatment effect estimates is zero; Test type: Superiority or Other; p = 0.407, ANCOVA; LS Mean Difference = -0.6, 90% CI 2-sided [-1.8 to 0.6], Standard Error of Mean 0.70
Statistical Analysis 36: Comparison: PF-06372865 2.5 mg (Stage 1) vs PF-06372865 7.5 mg (Stage 1) vs PF-06372865 2.5 mg (Stage 2) vs PF-06372865 7.5 mg (Stage 2); (PF-06372865 7.5 mg - PF-06372865 2.5 mg). Family Sub-Scale Score (Combined Stage 1 and Stage 2): The ANCOVA model included change from baseline as dependent variable, and treatment and baseline in the model. Baseline for Stage 1 is Day 1 and baseline for Stage 2 is Week 4 (Day 28). The estimates from Stage 1 and the Stage 2 were combined together using a weighted mean (weight=0.5) and assuming the covariance between the two treatment effect estimates is zero; Test type: Superiority or Other; p = 0.412, ANCOVA; LS Mean Difference = 0.6, 90% CI 2-sided [-0.6 to 1.7], Standard Error of Mean 0.66

7. Secondary Outcome: Change From Baseline in Hamilton Anxiety Rating Scale (HAM-A) Total Scores at Week 1, Week 2 and Week 3: Stage 1
Description: as for outcome 1
Time Frame: Week 1, 2, 3
Population: Stage 1 full analysis set: All randomized participants who received at least 1 dose of study treatment. Here, 'n' signifies those participants who were evaluable at specified time point for each arm, respectively.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (Stage 1) | PF-06372865 2.5 mg (Stage 1) | PF-06372865 7.5 mg (Stage 1)
Number analyzed (Participants) | 45 | 24 | 21
units on a scale
  Week 1 (n= 41,24,21) | -6.0 (0.84) | -5.3 (1.09) | -5.7 (1.18)
  Week 2 (n= 39,23,21) | -6.9 (1.05) | -6.3 (1.37) | -7.7 (1.45)
  Week 3 (n= 39,22,21) | -10.2 (1.00) | -8.6 (1.32) | -9.2 (1.38)
Statistical Analysis 1: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1); (PF-06372865 7.5 mg - Placebo). Week 1: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 1 was Day 1; Test type: Superiority or Other; p = 0.856, Mixed-Effects Model Repeated Measure; Least Squares Mean Difference = 0.3, 90% CI 2-sided [-2.2 to 2.7], Standard Error of Mean 1.45
Statistical Analysis 2: Comparison: Placebo (Stage 1) vs PF-06372865 2.5 mg (Stage 1); (PF-06372865 2.5 mg - Placebo). Week 1: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 1 was Day 1; Test type: Superiority or Other; p = 0.647, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.6, 90% CI 2-sided [-1.7 to 2.9], Standard Error of Mean 1.38
Statistical Analysis 3: Comparison: PF-06372865 2.5 mg (Stage 1) vs PF-06372865 7.5 mg (Stage 1); (PF-06372865 7.5 mg - PF-06372865 2.5 mg). Week 1: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 1 was Day 1; Test type: Superiority or Other; p = 0.817, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.4, 90% CI 2-sided [-3.0 to 2.3], Standard Error of Mean 1.60
Statistical Analysis 4: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1); (PF-06372865 7.5 mg - Placebo). Week 2: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 1 was Day 1; Test type: Superiority or Other; p = 0.670, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.8, 90% CI 2-sided [-3.8 to 2.2], Standard Error of Mean 1.81
Statistical Analysis 5: Comparison: Placebo (Stage 1) vs PF-06372865 2.5 mg (Stage 1); (PF-06372865 2.5 mg - Placebo). Week 2: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 1 was Day 1; Test type: Superiority or Other; p = 0.736, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.6, 90% CI 2-sided [-2.3 to 3.5], Standard Error of Mean 1.74
Statistical Analysis 6: Comparison: PF-06372865 2.5 mg (Stage 1) vs PF-06372865 7.5 mg (Stage 1); (PF-06372865 7.5 mg - PF-06372865 2.5 mg). Week 2: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 1 was Day 1; Test type: Superiority or Other; p = 0.496, Mixed-Effects Model Repeated Measure; LS Mean Difference = -1.4, 90% CI 2-sided [-4.7 to 2.0], Standard Error of Mean 1.99
Statistical Analysis 7: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1); (PF-06372865 7.5 mg - Placebo). Week 3: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 1 was Day 1; Test type: Superiority or Other; p = 0.575, Mixed-Effects Model Repeated Measure; LS Mean Difference = 1.0, 90% CI 2-sided [-1.9 to 3.8], Standard Error of Mean 1.72
Statistical Analysis 8: Comparison: Placebo (Stage 1) vs PF-06372865 2.5 mg (Stage 1); (PF-06372865 2.5 mg - Placebo). Week 3: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 1 was Day 1; Test type: Superiority or Other; p = 0.362, Mixed-Effects Model Repeated Measure; LS Mean Difference = 1.5, 90% CI 2-sided [-1.2 to 4.3], Standard Error of Mean 1.67
Statistical Analysis 9: Comparison: PF-06372865 2.5 mg (Stage 1) vs PF-06372865 7.5 mg (Stage 1); (PF-06372865 7.5 mg - PF-06372865 2.5 mg). Week 3: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 1 was Day 1; Test type: Superiority or Other; p = 0.771, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.6, 90% CI 2-sided [-3.7 to 2.6], Standard Error of Mean 1.90

8. Secondary Outcome: Percentage of Responders of Total Hamilton Anxiety Rating Scale (HAM-A): Stage 1 and Stage 2
Description: A responder was defined as a participant with >= to 50 percent decrease in their total HAM-A score from baseline to the last week in the stage (Week 4 in Stage 1, Week 8 in Stage 2). The HAM-A scale was a clinician rated interview scale designed to measure the signs and symptoms of anxiety. It had 14-items to rate the intensity of psychic and somatic anxiety on a 5-point severity scale. Each item ranging from 0 (not present) to 4 (very severe) were summed up to give a total possible score of 0 (not present) to 56 (very severe), where lower scores indicates less anxiety. Percentage of responders of total HMA scale were reported.
Time Frame: Stage 1: Week 4, Stage 2: Week 8
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Stage 1) | PF-06372865 2.5 mg (Stage 1) | PF-06372865 7.5 mg (Stage 1) | Placebo (Stage 2) | PF-06372865 2.5 mg (Stage 2) | PF-06372865 7.5 mg (Stage 2)
Number analyzed (Participants) | 45 | 24 | 21 | 6 | 8 | 8
percentage of participants | 33.33 | 25.00 | 28.57 | 16.67 | 25.00 | 12.50
Statistical Analysis 1: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1); (PF-06372865 7.5 mg - Placebo). Stage 1: Logistic regression model included treatment as fixed effect, and the baseline as covariate. Baseline for Stage 1 is Day 1 and for Stage 2 is Day 28; Test type: Superiority or Other; Regression, Logistic; Odds Ratio (OR) = 0.75, 90% CI 2-sided [0.45 to 1.26]
Statistical Analysis 2: Comparison: Placebo (Stage 1) vs PF-06372865 2.5 mg (Stage 1); (PF-06372865 2.5 mg - Placebo). Stage 1: Logistic regression model included treatment as fixed effect, and the baseline as covariate. Baseline for Stage 1 is Day 1 and for Stage 2 is Day 28; Test type: Superiority or Other; Regression, Logistic; Odds Ratio (OR) = 0.60, 90% CI 2-sided [0.23 to 1.54]
Statistical Analysis 3: Comparison: PF-06372865 2.5 mg (Stage 1) vs PF-06372865 7.5 mg (Stage 1); (PF-06372865 7.5 mg - PF-06372865 2.5 mg). Stage 1: Logistic regression model included treatment as fixed effect, and the baseline as covariate. Baseline for Stage 1 is Day 1 and for Stage 2 is Day 28; Test type: Superiority or Other; Regression, Logistic; Odds Ratio (OR) = 1.26, 90% CI 2-sided [0.69 to 2.32]
Statistical Analysis 4: Comparison: Placebo (Stage 2) vs PF-06372865 7.5 mg (Stage 2); (PF-06372865 7.5 mg - Placebo). Stage 2: Logistic regression model included treatment as fixed effect, and the baseline as covariate. Baseline for Stage 1 is Day 1 and for Stage 2 is Day 28; Test type: Superiority or Other; Regression, Logistic; Odds Ratio (OR) = 1.24, 90% CI 2-sided [0.27 to 5.78]
Statistical Analysis 5: Comparison: Placebo (Stage 2) vs PF-06372865 2.5 mg (Stage 2); (PF-06372865 2.5 mg - Placebo). Stage 2: Logistic regression model included treatment as fixed effect, and the baseline as covariate. Baseline for Stage 1 is Day 1 and for Stage 2 is Day 28; Test type: Superiority or Other; Regression, Logistic; Odds Ratio, log = 2.13, 90% CI 2-sided [0.19 to 24.51]
Statistical Analysis 6: Comparison: PF-06372865 2.5 mg (Stage 2) vs PF-06372865 7.5 mg (Stage 2); (PF-06372865 7.5 mg - PF-06372865 2.5 mg). Stage 2: Logistic regression model included treatment as fixed effect, and the baseline as covariate. Baseline for Stage 1 is Day 1 and for Stage 2 is Day 28; Test type: Superiority or Other; Regression, Logistic; Odds Ratio (OR) = 0.58, 90% CI 2-sided [0.16 to 2.09]

9. Secondary Outcome: Change From Baseline in Clinical Global Impression - Improvement (CGI-I) Scale Score at Week 1, 2, 3, 4 in Stage 1 and Week 5, 6, 7, 8 in Stage 2
Description: CGI-I was a 7-point clinician rated scale ranging from 1 (very much improved) to 7 (very much worse). Improvement was defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved), 4 (no change), 5 (minimally worse), 6 (much worse) or 7 (very much worse) on the scale. Higher score indicated more affected. Change is equal to score at observation minus score at baseline.
Time Frame: Stage 1 (S1): Baseline (Day 1), Week 1 (W1), 2 (W2), 3 (W3), 4 (W4) and Stage 2 (S2): Baseline (Day 28), Week 5 (W5), 6 (W6), 7 (W7), 8 (W8)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Stage 1) | PF-06372865 2.5 mg (Stage 1) | PF-06372865 7.5 mg (Stage 1) | Placebo (Stage 2) | PF-06372865 2.5 mg (Stage 2) | PF-06372865 7.5 mg (Stage 2)
Number analyzed (Participants) | 45 | 24 | 21 | 6 | 8 | 8
units on a scale
  Baseline : S1, S2 (n=45,23,21,6,8,8) | 3.8 (0.53) | 3.8 (0.74) | 3.9 (0.36) | 3.5 (0.55) | 3.3 (0.71) | 3.0 (0.76)
  Change at S1: W1, S2: W5 (n=41,23,21,6,8,8) | -0.4 (0.89) | -0.6 (1.04) | -0.5 (0.87) | -0.2 (0.98) | -0.5 (1.20) | 0.3 (0.46)
  Change at S1: W2, S2: W6 (n=39,22,21,6,8,8) | -0.6 (0.91) | -0.7 (1.17) | -0.9 (1.11) | -0.5 (1.22) | -0.3 (1.16) | 0.1 (0.64)
  Change at S1: W3, S2: W7 (n=39,21,21,6,8,7) | -1.0 (0.99) | -0.9 (1.20) | -1.1 (1.01) | -0.7 (1.03) | -0.8 (1.16) | 0.0 (0.58)
  Change at S1: W4, S2: W8 (n=40,21,20,6,8,7) | -1.1 (1.06) | -1.0 (1.24) | -1.1 (1.05) | -0.5 (1.38) | -1.0 (1.20) | -0.3 (0.76)
Statistical Analysis 1: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1); (PF-06372865 7.5 mg - Placebo). Week 1: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 1 was Day 1 and baseline for Stage 2 was Week 4 (Day 28); Test type: Superiority or Other; p = 0.801, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.1, 90% CI 2-sided [-0.4 to 0.3], Standard Error of Mean 0.21
Statistical Analysis 2: Comparison: Placebo (Stage 1) vs PF-06372865 2.5 mg (Stage 1); (PF-06372865 2.5 mg - Placebo). Week 1: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 1 was Day 1 and baseline for Stage 2 was Week 4 (Day 28); Test type: Superiority or Other; p = 0.416, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.2, 90% CI 2-sided [-0.5 to 0.2], Standard Error of Mean 0.20
Statistical Analysis 3: Comparison: PF-06372865 2.5 mg (Stage 1) vs PF-06372865 7.5 mg (Stage 1); (PF-06372865 7.5 mg - PF-06372865 2.5 mg). Week 1: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 1 was Day 1 and baseline for Stage 2 was Week 4 (Day 28); Test type: Superiority or Other; p = 0.634, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.1, 90% CI 2-sided [-0.3 to 0.5], Standard Error of Mean 0.23
Statistical Analysis 4: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1); (PF-06372865 7.5 mg - Placebo). Week 2: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 1 was Day 1 and baseline for Stage 2 was Week 4 (Day 28); Test type: Superiority or Other; p = 0.470, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.2, 90% CI 2-sided [-0.6 to 0.2], Standard Error of Mean 0.24
Statistical Analysis 5: Comparison: Placebo (Stage 1) vs PF-06372865 2.5 mg (Stage 1); (PF-06372865 2.5 mg - Placebo). Week 2: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 1 was Day 1 and baseline for Stage 2 was Week 4 (Day 28); Test type: Superiority or Other; p = 0.683, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.1, 90% CI 2-sided [-0.5 to 0.3], Standard Error of Mean 0.24
Statistical Analysis 6: Comparison: PF-06372865 2.5 mg (Stage 1) vs PF-06372865 7.5 mg (Stage 1); (PF-06372865 7.5 mg - PF-06372865 2.5 mg). Week 2: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 1 was Day 1 and baseline for Stage 2 was Week 4 (Day 28); Test type: Superiority or Other; p = 0.775, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.1, 90% CI 2-sided [-0.5 to 0.4], Standard Error of Mean 0.27
Statistical Analysis 7: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1); (PF-06372865 7.5 mg - Placebo). Week 3: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 1 was Day 1 and baseline for Stage 2 was Week 4 (Day 28); Test type: Superiority or Other; p = 0.848, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.0, 90% CI 2-sided [-0.4 to 0.3], Standard Error of Mean 0.24
Statistical Analysis 8: Comparison: Placebo (Stage 1) vs PF-06372865 2.5 mg (Stage 1); (PF-06372865 2.5 mg - Placebo). Week 3: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 1 was Day 1 and baseline for Stage 2 was Week 4 (Day 28); Test type: Superiority or Other; p = 0.490, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.2, 90% CI 2-sided [-0.2 to 0.6], Standard Error of Mean 0.23
Statistical Analysis 9: Comparison: PF-06372865 2.5 mg (Stage 1) vs PF-06372865 7.5 mg (Stage 1); (PF-06372865 7.5 mg - PF-06372865 2.5 mg). Week 3: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 1 was Day 1 and baseline for Stage 2 was Week 4 (Day 28); Test type: Superiority or Other; p = 0.433, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.2, 90% CI 2-sided [-0.7 to 0.2], Standard Error of Mean 0.27
Statistical Analysis 10: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1); (PF-06372865 7.5 mg - Placebo). Week 4: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 1 was Day 1 and baseline for Stage 2 was Week 4 (Day 28); Test type: Superiority or Other; p = 0.796, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.1, 90% CI 2-sided [-0.4 to 0.5], Standard Error of Mean 0.25
Statistical Analysis 11: Comparison: Placebo (Stage 1) vs PF-06372865 2.5 mg (Stage 1); (PF-06372865 2.5 mg - Placebo). Week 4: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 1 was Day 1 and baseline for Stage 2 was Week 4 (Day 28); Test type: Superiority or Other; p = 0.624, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.1, 90% CI 2-sided [-0.3 to 0.5], Standard Error of Mean 0.25
Statistical Analysis 12: Comparison: PF-06372865 2.5 mg (Stage 1) vs PF-06372865 7.5 mg (Stage 1); (PF-06372865 7.5 mg - PF-06372865 2.5 mg). Week 4: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 1 was Day 1 and baseline for Stage 2 was Week 4 (Day 28); Test type: Superiority or Other; p = 0.844, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.1, 90% CI 2-sided [-0.5 to 0.4], Standard Error of Mean 0.28
Statistical Analysis 13: Comparison: Placebo (Stage 2) vs PF-06372865 7.5 mg (Stage 2); (PF-06372865 7.5 mg - Placebo). Week 5: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 1 was Day 1 and baseline for Stage 2 was Week 4 (Day 28); Test type: Superiority or Other; p = 0.743, LS Mean Difference; LS Mean Difference = 0.2, 90% CI 2-sided [-0.7 to 1.0], Standard Error of Mean 0.50
Statistical Analysis 14: Comparison: Placebo (Stage 2) vs PF-06372865 2.5 mg (Stage 2); (PF-06372865 2.5 mg - Placebo). Week 5: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 1 was Day 1 and baseline for Stage 2 was Week 4 (Day 28); Test type: Superiority or Other; p = 0.356, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.5, 90% CI 2-sided [-1.3 to 0.4], Standard Error of Mean 0.48
Statistical Analysis 15: Comparison: PF-06372865 2.5 mg (Stage 2) vs PF-06372865 7.5 mg (Stage 2); (PF-06372865 7.5 mg - PF-06372865 2.5 mg). Week 5: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 1 was Day 1 and baseline for Stage 2 was Week 4 (Day 28); Test type: Superiority or Other; p = 0.180, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.6, 90% CI 2-sided [-0.2 to 1.4], Standard Error of Mean 0.45
Statistical Analysis 16: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1); (PF-06372865 7.5 mg - Placebo). Week 6: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 1 was Day 1 and baseline for Stage 2 was Week 4 (Day 28); Test type: Superiority or Other; p = 0.589, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.3, 90% CI 2-sided [-0.6 to 1.2], Standard Error of Mean 0.53
Statistical Analysis 17: Comparison: Placebo (Stage 2) vs PF-06372865 2.5 mg (Stage 2); (PF-06372865 2.5 mg - Placebo). Week 6: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 1 was Day 1 and baseline for Stage 2 was Week 4 (Day 28); Test type: Superiority or Other; p = 0.873, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.1, 90% CI 2-sided [-0.8 to 1.0], Standard Error of Mean 0.51
Statistical Analysis 18: Comparison: PF-06372865 2.5 mg (Stage 2) vs PF-06372865 7.5 mg (Stage 2); (PF-06372865 7.5 mg - PF-06372865 2.5 mg). Week 6: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 1 was Day 1 and baseline for Stage 2 was Week 4 (Day 28); Test type: Superiority or Other; p = 0.667, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.2, 90% CI 2-sided [-0.6 to 1.0], Standard Error of Mean 0.48
Statistical Analysis 19: Comparison: Placebo (Stage 2) vs PF-06372865 7.5 mg (Stage 2); (PF-06372865 7.5 mg - Placebo). Week 7: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 1 was Day 1 and baseline for Stage 2 was Week 4 (Day 28); Test type: Superiority or Other; p = 0.548, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.3, 90% CI 2-sided [-0.5 to 1.1], Standard Error of Mean 0.47
Statistical Analysis 20: Comparison: Placebo (Stage 2) vs PF-06372865 2.5 mg (Stage 2); (PF-06372865 2.5 mg - Placebo). Week 7: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 1 was Day 1 and baseline for Stage 2 was Week 4 (Day 28); Test type: Superiority or Other; p = 0.567, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.3, 90% CI 2-sided [-1.0 to 0.5], Standard Error of Mean 0.45
Statistical Analysis 21: Comparison: PF-06372865 2.5 mg (Stage 2) vs PF-06372865 7.5 mg (Stage 2); (PF-06372865 7.5 mg - PF-06372865 2.5 mg). Week 7: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 1 was Day 1 and baseline for Stage 2 was Week 4 (Day 28); Test type: Superiority or Other; p = 0.208, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.6, 90% CI 2-sided [-0.2 to 1.3], Standard Error of Mean 0.42
Statistical Analysis 22: Comparison: Placebo (Stage 2) vs PF-06372865 7.5 mg (Stage 2); (PF-06372865 7.5 mg - Placebo). Week 8: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 1 was Day 1 and baseline for Stage 2 was Week 4 (Day 28); Test type: Superiority or Other; p = 0.858, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.1, 90% CI 2-sided [-1.2 to 0.9], Standard Error of Mean 0.60
Statistical Analysis 23: Comparison: Placebo (Stage 2) vs PF-06372865 2.5 mg (Stage 2); (PF-06372865 2.5 mg - Placebo). Week 8: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 1 was Day 1 and baseline for Stage 2 was Week 4 (Day 28); Test type: Superiority or Other; p = 0.329, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.7, 90% CI 2-sided [-1.7 to 0.3], Standard Error of Mean 0.58
Statistical Analysis 24: Comparison: PF-06372865 2.5 mg (Stage 2) vs PF-06372865 7.5 mg (Stage 2); (PF-06372865 7.5 mg - PF-06372865 2.5 mg). Week 8: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 1 was Day 1 and baseline for Stage 2 was Week 4 (Day 28); Test type: Superiority or Other; p = 0.272, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.5, 90% CI 2-sided [-0.4 to 1.5], Standard Error of Mean 0.54
Statistical Analysis 25: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1) vs Placebo (Stage 2) vs PF-06372865 7.5 mg (Stage 2); (PF-06372865 7.5 mg - Placebo). Combined Stage 1 (Week 4) and Stage 2 (Week 8): Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect; Test type: Superiority or Other; p = 0.946, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.0, 90% CI 2-sided [-0.6 to 0.5], Standard Error of Mean 0.33
Statistical Analysis 26: Comparison: Placebo (Stage 1) vs PF-06372865 2.5 mg (Stage 1) vs Placebo (Stage 2) vs PF-06372865 2.5 mg (Stage 2); (PF-06372865 2.5 mg - Placebo). Combined Stage 1 (Week 4) and Stage 2 (Week 8): Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect; Test type: Superiority or Other; p = 0.407, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.3, 90% CI 2-sided [-0.8 to 0.3], Standard Error of Mean 0.31
Statistical Analysis 27: Comparison: PF-06372865 2.5 mg (Stage 1) vs PF-06372865 7.5 mg (Stage 1) vs PF-06372865 2.5 mg (Stage 2) vs PF-06372865 7.5 mg (Stage 2); (PF-06372865 7.5 mg - PF-06372865 2.5 mg). Combined Stage 1 (Week 4) and Stage 2 (Week 8): Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect; Test type: Superiority or Other; p = 0.436, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.2, 90% CI 2-sided [-0.3 to 0.8], Standard Error of Mean 0.31

10. Secondary Outcome: Change From Baseline in Clinical Global Impression -Severity (CGI-S) Scale Score at Week 1, 2, 3, 4 in Stage 1 and Week 5, 6, 7, 8 in Stage 2
Description: The CGI-S consisted of a single 7-point rating score of illness severity, was completed by a clinician. Raters selected one response based on the following question, "Considering your total clinical experience with that particular population, how mentally ill was your participant at that time?" Scores were: 1 (normal, not ill at all), 2 (borderline mentally ill), 3 (mildly ill), 4 (moderately ill), 5 (markedly ill) 6 (severely ill) or 7 (among the most severely ill participants). Higher scores indicate more severity.
Time Frame: as for outcome 9
Population: Full analysis set for Stage 1 and Placebo Non-Responder set for Stage 2. Here, number of participants analyzed (N) signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Stage 1) | PF-06372865 2.5 mg (Stage 1) | PF-06372865 7.5 mg (Stage 1) | Placebo (Stage 2) | PF-06372865 2.5 mg (Stage 2) | PF-06372865 7.5 mg (Stage 2)
Number analyzed (Participants) | 45 | 24 | 21 | 6 | 8 | 8
units on a scale
  Baseline: S1 and S2 (n=45,24,21,6,8,8) | 4.8 (0.63) | 4.6 (0.58) | 4.8 (0.54) | 4.5 (1.05) | 4.3 (0.89) | 4.0 (0.76)
  Change at S1: W1, S2: W5 (n=41,24,21,6,8,8) | -0.5 (0.78) | -0.5 (0.93) | -0.7 (0.72) | 0.0 (1.10) | -0.1 (0.99) | 0.0 (0.53)
  Change at S1: W2, S2: W6 (n=39,23,21,6,8,8) | -0.8 (0.90) | -0.7 (1.01) | -1.0 (1.07) | -0.5 (1.64) | 0.0 (0.93) | -0.1 (0.64)
  Change at S1: W3, S2: W7 (n=39,22,21,6,8,7) | -1.2 (1.12) | -1.0 (1.21) | -1.4 (0.98) | -0.8 (1.33) | -1.0 (0.93) | -0.3 (0.49)
  Change at S1: W4, S2: W8 (n=40,22,20,6,8,7) | -1.3 (1.16) | -1.0 (1.21) | -1.3 (1.08) | -0.5 (1.87) | -1.1 (0.83) | -0.6 (0.79)
Statistical Analysis 1: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1); (PF-06372865 7.5 mg - Placebo). Week 1: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect; Test type: Superiority or Other; p = 0.325, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.2, 90% CI 2-sided [-0.6 to 0.1], Standard Error of Mean 0.21
Statistical Analysis 2: Comparison: Placebo (Stage 1) vs PF-06372865 2.5 mg (Stage 1); [analysis description as in outcome 9, analysis 2]; Test type: Superiority or Other; p = 0.996, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.0, 90% CI 2-sided [-0.3 to 0.3], Standard Error of Mean 0.20
Statistical Analysis 3: Comparison: PF-06372865 2.5 mg (Stage 1) vs PF-06372865 7.5 mg (Stage 1); [analysis description as in outcome 9, analysis 3]; Test type: Superiority or Other; p = 0.377, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.2, 90% CI 2-sided [-0.6 to 0.2], Standard Error of Mean 0.24
Statistical Analysis 4: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1); [analysis description as in outcome 9, analysis 4]; Test type: Superiority or Other; p = 0.291, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.3, 90% CI 2-sided [-0.7 to 0.1], Standard Error of Mean 0.24
Statistical Analysis 5: Comparison: Placebo (Stage 1) vs PF-06372865 2.5 mg (Stage 1); [analysis description as in outcome 9, analysis 5]; Test type: Superiority or Other; p = 0.925, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.0, 90% CI 2-sided [-0.4 to 0.4], Standard Error of Mean 0.24
Statistical Analysis 6: Comparison: PF-06372865 2.5 mg (Stage 1) vs PF-06372865 7.5 mg (Stage 1); [analysis description as in outcome 9, analysis 6]; Test type: Superiority or Other; p = 0.390, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.2, 90% CI 2-sided [-0.7 to 0.2], Standard Error of Mean 0.27
Statistical Analysis 7: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1); [analysis description as in outcome 9, analysis 7]; Test type: Superiority or Other; p = 0.502, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.2, 90% CI 2-sided [-0.7 to 0.3], Standard Error of Mean 0.29
Statistical Analysis 8: Comparison: Placebo (Stage 1) vs PF-06372865 2.5 mg (Stage 1); [analysis description as in outcome 9, analysis 8]; Test type: Superiority or Other; p = 0.348, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.3, 90% CI 2-sided [-0.2 to 0.7], Standard Error of Mean 0.29
Statistical Analysis 9: Comparison: PF-06372865 2.5 mg (Stage 1) vs PF-06372865 7.5 mg (Stage 1); [analysis description as in outcome 9, analysis 9]; Test type: Superiority or Other; p = 0.160, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.5, 90% CI 2-sided [-1.0 to 0.1], Standard Error of Mean 0.33
Statistical Analysis 10: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1); [analysis description as in outcome 9, analysis 10]; Test type: Superiority or Other; p = 0.965, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.0, 90% CI 2-sided [-0.5 to 0.5], Standard Error of Mean 0.30
Statistical Analysis 11: Comparison: Placebo (Stage 1) vs PF-06372865 2.5 mg (Stage 1); [analysis description as in outcome 9, analysis 11]; Test type: Superiority or Other; p = 0.389, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.3, 90% CI 2-sided [-0.2 to 0.7], Standard Error of Mean 0.30
Statistical Analysis 12: Comparison: PF-06372865 2.5 mg (Stage 1) vs PF-06372865 7.5 mg (Stage 1); [analysis description as in outcome 9, analysis 12]; Test type: Superiority or Other; p = 0.433, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.3, 90% CI 2-sided [-0.8 to 0.3], Standard Error of Mean 0.34
Statistical Analysis 13: Comparison: Placebo (Stage 2) vs PF-06372865 7.5 mg (Stage 2); [analysis description as in outcome 9, analysis 13]; Test type: Superiority or Other; p = 0.940, LS Mean Difference; LS Mean Difference = -0.1, 90% CI 2-sided [-0.9 to 0.8], Standard Error of Mean 0.50
Statistical Analysis 14: Comparison: Placebo (Stage 2) vs PF-06372865 2.5 mg (Stage 2); [analysis description as in outcome 9, analysis 14]; Test type: Superiority or Other; p = 0.757, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.2, 90% CI 2-sided [-1.0 to 0.7], Standard Error of Mean 0.49
Statistical Analysis 15: Comparison: PF-06372865 2.5 mg (Stage 2) vs PF-06372865 7.5 mg (Stage 2); [analysis description as in outcome 9, analysis 15]; Test type: Superiority or Other; p = 0.836, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.1, 90% CI 2-sided [-0.7 to 0.9], Standard Error of Mean 0.46
Statistical Analysis 16: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1); [analysis description as in outcome 9, analysis 16]; Test type: Superiority or Other; p = 0.827, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.1, 90% CI 2-sided [-0.9 to 1.1], Standard Error of Mean 0.56
Statistical Analysis 17: Comparison: Placebo (Stage 2) vs PF-06372865 2.5 mg (Stage 2); [analysis description as in outcome 9, analysis 17]; Test type: Superiority or Other; p = 0.507, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.4, 90% CI 2-sided [-0.6 to 1.3], Standard Error of Mean 0.55
Statistical Analysis 18: Comparison: PF-06372865 2.5 mg (Stage 2) vs PF-06372865 7.5 mg (Stage 2); [analysis description as in outcome 9, analysis 18]; Test type: Superiority or Other; p = 0.632, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.3, 90% CI 2-sided [-1.1 to 0.6], Standard Error of Mean 0.51
Statistical Analysis 19: Comparison: Placebo (Stage 2) vs PF-06372865 7.5 mg (Stage 2); [analysis description as in outcome 9, analysis 19]; Test type: Superiority or Other; p = 0.442, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.4, 90% CI 2-sided [-0.5 to 1.3], Standard Error of Mean 0.51
Statistical Analysis 20: Comparison: Placebo (Stage 2) vs PF-06372865 2.5 mg (Stage 2); [analysis description as in outcome 9, analysis 20]; Test type: Superiority or Other; p = 0.643, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.2, 90% CI 2-sided [-1.1 to 0.6], Standard Error of Mean 0.50
Statistical Analysis 21: Comparison: PF-06372865 2.5 mg (Stage 2) vs PF-06372865 7.5 mg (Stage 2); [analysis description as in outcome 9, analysis 21]; Test type: Superiority or Other; p = 0.188, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.6, 90% CI 2-sided [-0.2 to 1.5], Standard Error of Mean 0.47
Statistical Analysis 22: Comparison: Placebo (Stage 2) vs PF-06372865 7.5 mg (Stage 2); [analysis description as in outcome 9, analysis 22]; Test type: Superiority or Other; p = 0.701, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.3, 90% CI 2-sided [-1.4 to 0.9], Standard Error of Mean 0.65
Statistical Analysis 23: Comparison: Placebo (Stage 2) vs PF-06372865 2.5 mg (Stage 2); [analysis description as in outcome 9, analysis 23]; Test type: Superiority or Other; p = 0.271, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.7, 90% CI 2-sided [-1.8 to 0.4], Standard Error of Mean 0.63
Statistical Analysis 24: Comparison: PF-06372865 2.5 mg (Stage 2) vs PF-06372865 7.5 mg (Stage 2); [analysis description as in outcome 9, analysis 24]; Test type: Superiority or Other; p = 0.445, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.5, 90% CI 2-sided [-0.6 to 1.5], Standard Error of Mean 0.60
Statistical Analysis 25: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1) vs Placebo (Stage 2) vs PF-06372865 7.5 mg (Stage 2); [analysis description as in outcome 9, analysis 25]; Test type: Superiority or Other; p = 0.714, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.1, 90% CI 2-sided [-0.8 to 0.5], Standard Error of Mean 0.36
Statistical Analysis 26: Comparison: Placebo (Stage 1) vs PF-06372865 2.5 mg (Stage 1) vs Placebo (Stage 2) vs PF-06372865 2.5 mg (Stage 2); [analysis description as in outcome 9, analysis 26]; Test type: Superiority or Other; p = 0.515, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.2, 90% CI 2-sided [-0.8 to 0.4], Standard Error of Mean 0.35
Statistical Analysis 27: Comparison: PF-06372865 2.5 mg (Stage 1) vs PF-06372865 7.5 mg (Stage 1) vs PF-06372865 2.5 mg (Stage 2) vs PF-06372865 7.5 mg (Stage 2); [analysis description as in outcome 9, analysis 27]; Test type: Superiority or Other; p = 0.778, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.1, 90% CI 2-sided [-0.5 to 0.7], Standard Error of Mean 0.34

11. Secondary Outcome: Plasma Concentration Versus Time Summary of PF-06372865: Stage 1
Description: Concentration versus time summary was calculated by setting concentration values below the lower limit of quantification (LLOQ =0.0100 nanogram per milliliter (ng/mL) to zero. Summary statistics were not to be presented if number of observations above lower limit of quantification (NALQ) = 0.
Time Frame: Pre-dose (0 hour), 2, 4, 10 hours post dose on Day 1 of Week 2, 3, 4
Population: Stage 1 full analysis set: All randomized participants who received at least 1 dose of study treatment. Participants who received PF-06372865 2.5 mg or PF-06372865 7.5 mg were evaluable for this measure. Here,'n' signifies those participants who were evaluable at specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-06372865 2.5 mg (Stage 1) | PF-06372865 7.5 mg (Stage 1)
Number analyzed (Participants) | 24 | 21
ng/mL
  Week 2 : 0 Hour (n= 12, 10) | 10.89 (7.1367) | 64.73 (58.463)
  Week 2 : 2 Hour (n= 13, 10) | 20.76 (10.060) | 113.8 (55.517)
  Week 2 : 4 Hour (n= 5, 8) | 16.07 (18.541) | 77.75 (65.594)
  Week 2 : 10 Hour (n= 5, 9) | 17.41 (14.951) | 66.60 (53.888)
  Week 3 : 0 Hour (n= 6, 5) | 11.62 (10.440) | 33.44 (34.409)
  Week 3 : 2 Hour (n= 6, 4) | 16.42 (13.626) | 54.02 (54.091)
  Week 3 : 4 Hour (n= 10, 9) | 22.20 (19.110) | 81.58 (54.133)
  Week 3 : 10 Hour (n= 10, 9) | 19.40 (13.880) | 73.31 (57.082)
  Week 4 : 0 Hour (n= 7, 9) | 14.36 (18.770) | 27.15 (20.840)
  Week 4 : 2 Hour (n= 8, 10) | 26.32 (20.328) | 61.98 (21.457)
  Week 4 : 4 Hour (n= 11, 5) | 29.58 (12.398) | 79.00 (69.914)
  Week 4 : 10 Hour (n= 10, 5) | 28.48 (11.550) | 78.60 (81.529)

12. Secondary Outcome: Plasma Concentration Versus Time Summary of PF-06372865: Stage 2
Description: Concentration versus time summary was calculated by setting concentration values below the lower limit of quantification (LLOQ =0.0100 ng/mL) to zero. Summary statistics were not to be presented if number of observations above lower limit of quantification (NALQ) =0.
Time Frame: Pre-dose (0 hour), 2, 4, 10 hours post dose on Day 1 of Week 6, 7, 8
Population: Placebo Non-Responder set for Stage 2. Participants who received PF-06372865 2.5 mg or PF-06372865 7.5 mg were evaluable for this measure. Here,'n' signifies those participants who were evaluable at specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-06372865 2.5 mg (Stage 2) | PF-06372865 7.5 mg (Stage 2)
Number analyzed (Participants) | 8 | 8
ng/mL
  Week 6 : 0 Hour (n= 3, 2) | 23.12 (22.644) | 35.67 (31.015)
  Week 6 : 2 Hour (n= 5, 3) | 24.62 (16.959) | 59.40 (46.218)
  Week 6 : 4 Hour (n= 2, 3) | 16.83 (19.459) | 75.98 (60.380)
  Week 6 : 10 Hour (n= 2, 3) | 14.00 (16.191) | 66.43 (52.402)
  Week 7 : 0 Hour (n= 3, 3) | 25.88 (20.591) | 17.54 (9.7180)
  Week 7 : 2 Hour (n= 4, 2) | 24.54 (17.913) | 16.40 (14.262)
  Week 7 : 4 Hour (n= 3, 4) | 34.80 (44.089) | 57.28 (38.837)
  Week 7 : 10 Hour (n= 3, 4) | 33.54 (38.779) | 64.45 (22.420)
  Week 8 : 0 Hour (n= 3, 5) | 25.18 (17.783) | 32.73 (25.175)
  Week 8 : 2 Hour (n= 4, 6) | 34.55 (14.856) | 48.83 (39.032)
  Week 8 : 4 Hour (n= 4, 3) | 13.54 (15.435) | 13.54 (15.435)
  Week 8 : 10 Hour (n= 3, 2) | 14.00 (15.880) | 14.00 (15.880)

13. Secondary Outcome: Change From Baseline in the Hamilton Anxiety Rating Scale (HAM-A): Psychic Subscale Score at Week 1, 2, 3, 4, 5, 6, 7, 8
Description: The HAM-A scale was a clinician interview-administered scale designed to measure the signs and symptoms of anxiety. It had 14-items to rate the intensity of psychic and somatic anxiety on a 5-point severity scale. Psychic subscale of the HAM-A was the sum of 7 items. Each item ranging from 0 (not present) to 4 (very severe) were summed up to give a total possible score of 0 (not present) to 28 (very severe), where lower scores indicates less anxiety.
Time Frame: as for outcome 9
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Stage 1) | PF-06372865 2.5 mg (Stage 1) | PF-06372865 7.5 mg (Stage 1) | Placebo (Stage 2) | PF-06372865 2.5 mg (Stage 2) | PF-06372865 7.5 mg (Stage 2)
Number analyzed (Participants) | 45 | 24 | 21 | 6 | 8 | 8
units on a scale
  Baseline: S1 and S2 (n=45,24,21,6,8,8) | 16.5 (2.23) | 15.2 (2.36) | 16.1 (1.77) | 15.5 (2.88) | 13.0 (4.54) | 12.9 (3.87)
  Change at S1: W1, S2: W5 (n=41,24, 21,6,8,8) | -2.8 (3.87) | -2.7 (3.42) | -3.2 (2.87) | -0.3 (2.88) | -0.6 (2.83) | 0.3 (1.28)
  Change at S1: W2, S2: W6 (n=39,23,21,6,8,8) | -3.8 (3.92) | -3.4 (4.97) | -4.6 (4.35) | -0.8 (2.86) | 0.4 (2.97) | -0.6 (2.20)
  Change at S1: W3, S2: W7 (n=39,22,21,6,8,7) | -5.3 (4.21) | -4.4 (4.53) | -5.4 (3.63) | -1.7 (2.42) | -2.3 (3.28) | -0.7 (1.80)
  Change at S1: W4, S2: W8 (n=40,22,20,6,8,7) | -5.9 (4.63) | -4.0 (5.19) | -5.8 (3.89) | -2.5 (3.56) | -3.9 (3.27) | -1.6 (3.05)
Statistical Analysis 1: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1); [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.562, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.5, 90% CI 2-sided [-2.1 to 1.0], Standard Error of Mean 0.93
Statistical Analysis 2: Comparison: Placebo (Stage 1) vs PF-06372865 2.5 mg (Stage 1); [analysis description as in outcome 9, analysis 2]; Test type: Superiority or Other; p = 0.708, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.3, 90% CI 2-sided [-1.9 to 1.2], Standard Error of Mean 0.92
Statistical Analysis 3: Comparison: PF-06372865 2.5 mg (Stage 1) vs PF-06372865 7.5 mg (Stage 1); [analysis description as in outcome 9, analysis 3]; Test type: Superiority or Other; p = 0.852, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.2, 90% CI 2-sided [-1.9 to 1.5], Standard Error of Mean 1.05
Statistical Analysis 4: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1); [analysis description as in outcome 9, analysis 4]; Test type: Superiority or Other; p = 0.347, Mixed-Effects Model Repeated Measure; LS Mean Difference = -1.1, 90% CI 2-sided [-3.0 to 0.8], Standard Error of Mean 1.14
Statistical Analysis 5: Comparison: Placebo (Stage 1) vs PF-06372865 2.5 mg (Stage 1); [analysis description as in outcome 9, analysis 5]; Test type: Superiority or Other; p = 0.759, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.4, 90% CI 2-sided [-2.2 to 1.5], Standard Error of Mean 1.14
Statistical Analysis 6: Comparison: PF-06372865 2.5 mg (Stage 1) vs PF-06372865 7.5 mg (Stage 1); [analysis description as in outcome 9, analysis 6]; Test type: Superiority or Other; p = 0.574, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.7, 90% CI 2-sided [-2.9 to 1.4], Standard Error of Mean 1.28
Statistical Analysis 7: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1); [analysis description as in outcome 9, analysis 7]; Test type: Superiority or Other; p = 0.831, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.2, 90% CI 2-sided [-2.1 to 1.6], Standard Error of Mean 1.09
Statistical Analysis 8: Comparison: Placebo (Stage 1) vs PF-06372865 2.5 mg (Stage 1); [analysis description as in outcome 9, analysis 8]; Test type: Superiority or Other; p = 0.705, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.4, 90% CI 2-sided [-1.4 to 2.3], Standard Error of Mean 1.10
Statistical Analysis 9: Comparison: PF-06372865 2.5 mg (Stage 1) vs PF-06372865 7.5 mg (Stage 1); [analysis description as in outcome 9, analysis 9]; Test type: Superiority or Other; p = 0.600, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.7, 90% CI 2-sided [-2.7 to 1.4], Standard Error of Mean 1.24
Statistical Analysis 10: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1); [analysis description as in outcome 9, analysis 10]; Test type: Superiority or Other; p = 0.848, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.2, 90% CI 2-sided [-2.3 to 1.8], Standard Error of Mean 1.23
Statistical Analysis 11: Comparison: Placebo (Stage 1) vs PF-06372865 2.5 mg (Stage 1); [analysis description as in outcome 9, analysis 11]; Test type: Superiority or Other; p = 0.237, Mixed-Effects Model Repeated Measure; LS Mean Difference = 1.5, 90% CI 2-sided [-0.6 to 3.5], Standard Error of Mean 1.24
Statistical Analysis 12: Comparison: PF-06372865 2.5 mg (Stage 1) vs PF-06372865 7.5 mg (Stage 1); [analysis description as in outcome 9, analysis 12]; Test type: Superiority or Other; p = 0.224, Mixed-Effects Model Repeated Measure; LS Mean Difference = -1.7, 90% CI 2-sided [-4.0 to 0.6], Standard Error of Mean 1.40
Statistical Analysis 13: Comparison: Placebo (Stage 2) vs PF-06372865 7.5 mg (Stage 2); [analysis description as in outcome 9, analysis 13]; Test type: Superiority or Other; p = 0.747, LS Mean Difference; LS Mean Difference = 0.4, 90% CI 2-sided [-1.9 to 2.8], Standard Error of Mean 1.38
Statistical Analysis 14: Comparison: Placebo (Stage 2) vs PF-06372865 2.5 mg (Stage 2); (PF-06372865 2.5 mg - Placebo). Week 5: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect. Baseline for Stage 1 was Day 1 and baseline for Stage 2 was Week 4 (Day 28). Baseline for Stage 1 was Day 1 and baseline for Stage 2 was Week 4 (Day 28); Test type: Superiority or Other; p = 0.764, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.4, 90% CI 2-sided [-2.8 to 2.0], Standard Error of Mean 1.37
Statistical Analysis 15: Comparison: PF-06372865 2.5 mg (Stage 2) vs PF-06372865 7.5 mg (Stage 2); [analysis description as in outcome 9, analysis 15]; Test type: Superiority or Other; p = 0.487, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.9, 90% CI 2-sided [-1.3 to 3.0], Standard Error of Mean 1.22
Statistical Analysis 16: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1); [analysis description as in outcome 9, analysis 16]; Test type: Superiority or Other; p = 0.744, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.5, 90% CI 2-sided [-2.1 to 3.2], Standard Error of Mean 1.53
Statistical Analysis 17: Comparison: Placebo (Stage 2) vs PF-06372865 2.5 mg (Stage 2); [analysis description as in outcome 9, analysis 17]; Test type: Superiority or Other; p = 0.340, Mixed-Effects Model Repeated Measure; LS Mean Difference = 1.5, 90% CI 2-sided [-1.1 to 4.1], Standard Error of Mean 1.52
Statistical Analysis 18: Comparison: PF-06372865 2.5 mg (Stage 2) vs PF-06372865 7.5 mg (Stage 2); [analysis description as in outcome 9, analysis 18]; Test type: Superiority or Other; p = 0.477, Mixed-Effects Model Repeated Measure; LS Mean Difference = -1.0, 90% CI 2-sided [-3.3 to 1.4], Standard Error of Mean 1.36
Statistical Analysis 19: Comparison: Placebo (Stage 2) vs PF-06372865 7.5 mg (Stage 2); [analysis description as in outcome 9, analysis 19]; Test type: Superiority or Other; p = 0.482, Mixed-Effects Model Repeated Measure; LS Mean Difference = 1.1, 90% CI 2-sided [-1.5 to 3.7], Standard Error of Mean 1.51
Statistical Analysis 20: Comparison: Placebo (Stage 2) vs PF-06372865 2.5 mg (Stage 2); [analysis description as in outcome 9, analysis 20]; Test type: Superiority or Other; p = 0.719, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.5, 90% CI 2-sided [-3.1 to 2.0], Standard Error of Mean 1.49
Statistical Analysis 21: Comparison: PF-06372865 2.5 mg (Stage 2) vs PF-06372865 7.5 mg (Stage 2); [analysis description as in outcome 9, analysis 21]; Test type: Superiority or Other; p = 0.245, Mixed-Effects Model Repeated Measure; LS Mean Difference = 1.6, 90% CI 2-sided [-0.7 to 4.0], Standard Error of Mean 1.36
Statistical Analysis 22: Comparison: Placebo (Stage 2) vs PF-06372865 7.5 mg (Stage 2); [analysis description as in outcome 9, analysis 22]; Test type: Superiority or Other; p = 0.586, Mixed-Effects Model Repeated Measure; LS Mean Difference = 1.1, 90% CI 2-sided [-2.3 to 4.4], Standard Error of Mean 1.93
Statistical Analysis 23: Comparison: Placebo (Stage 2) vs PF-06372865 2.5 mg (Stage 2); [analysis description as in outcome 9, analysis 23]; Test type: Superiority or Other; p = 0.440, Mixed-Effects Model Repeated Measure; LS Mean Difference = -1.5, 90% CI 2-sided [-4.8 to 1.8], Standard Error of Mean 1.90
Statistical Analysis 24: Comparison: PF-06372865 2.5 mg (Stage 2) vs PF-06372865 7.5 mg (Stage 2); [analysis description as in outcome 9, analysis 24]; Test type: Superiority or Other; p = 0.159, Mixed-Effects Model Repeated Measure; LS Mean Difference = 2.6, 90% CI 2-sided [-0.5 to 5.6], Standard Error of Mean 1.75
Statistical Analysis 25: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1) vs Placebo (Stage 2) vs PF-06372865 7.5 mg (Stage 2); (PF-06372865 7.5 mg - Placebo). Combined Stage 1 and Stage 2: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect; Test type: Superiority or Other; p = 0.720, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.4, 90% CI 2-sided [-1.6 to 2.4], Standard Error of Mean 1.15
Statistical Analysis 26: Comparison: Placebo (Stage 1) vs PF-06372865 2.5 mg (Stage 1) vs Placebo (Stage 2) vs PF-06372865 2.5 mg (Stage 2); (PF-06372865 2.5 mg - Placebo). Combined Stage 1 and Stage 2: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect; Test type: Superiority or Other; p = 0.991, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.0, 90% CI 2-sided [-2.0 to 1.9], Standard Error of Mean 1.13
Statistical Analysis 27: Comparison: PF-06372865 2.5 mg (Stage 1) vs PF-06372865 7.5 mg (Stage 1) vs PF-06372865 2.5 mg (Stage 2) vs PF-06372865 7.5 mg (Stage 2); (PF-06372865 7.5 mg - PF-06372865 2.5 mg). Combined Stage 1 and Stage 2: Repeated measures model included week*treatment and baseline*week interaction as fixed effects, week repeated in each participant as repeated effect; Test type: Superiority or Other; p = 0.704, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.4, 90% CI 2-sided [-1.5 to 2.4], Standard Error of Mean 1.12

14. Secondary Outcome: Change From Baseline in the Hamilton Anxiety Rating Scale (HAM-A): Somatic Subscale Score at Week 1, 2, 3, 4, 5, 6, 7, 8
Description: The HAM-A scale was a clinician interview-administered scale designed to measure the signs and symptoms of anxiety. It had 14-items to rate the intensity of psychic and somatic anxiety on a 5-point severity scale. Somatic subscale of the HAM-A was the sum of 7 items. Each item ranging from 0 (not present) to 4 (very severe) were summed up to give a total possible score of 0 (not present) to 28 (very severe), where lower scores indicates less anxiety.
Time Frame: as for outcome 9
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Stage 1) | PF-06372865 2.5 mg (Stage 1) | PF-06372865 7.5 mg (Stage 1) | Placebo (Stage 2) | PF-06372865 2.5 mg (Stage 2) | PF-06372865 7.5 mg (Stage 2)
Number analyzed (Participants) | 45 | 24 | 21 | 6 | 8 | 8
units on a scale
  Baseline: S1 and S2 (n=45,24,21,6,8,8) | 11.5 (3.76) | 11.5 (3.15) | 10.0 (4.01) | 10.7 (5.20) | 9.5 (2.98) | 9.6 (3.34)
  Change at S1: W1, S2: W5 (n=41,24, 21,6,8,8) | -3.2 (3.37) | -2.6 (2.90) | -2.4 (2.77) | -0.3 (3.78) | -0.8 (2.60) | 0.4 (2.07)
  Change at S1: W2, S2: W6 (n=39,23,21,6,8,8) | -3.2 (3.09) | -2.8 (2.24) | -2.9 (4.27) | -2.7 (4.68) | -1.1 (2.03) | -0.5 (3.51)
  Change at S1: W3, S2: W7 (n=39,22,21,6,8,7) | -4.9 (3.63) | -4.1 (3.19) | -3.6 (3.47) | -2.8 (3.66) | -2.3 (2.82) | -1.3 (3.50)
  Change at S1: W4, S2: W8 (n=40,22,20,6,8,7) | -4.8 (4.62) | -3.7 (3.27) | -3.8 (3.49) | -2.0 (5.62) | -3.1 (3.14) | -2.0 (4.08)
Statistical Analysis 1: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1); [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.539, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.5, 90% CI 2-sided [-0.9 to 1.9], Standard Error of Mean 0.82
Statistical Analysis 2: Comparison: Placebo (Stage 1) vs PF-06372865 2.5 mg (Stage 1); [analysis description as in outcome 9, analysis 2]; Test type: Superiority or Other; p = 0.439, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.6, 90% CI 2-sided [-0.7 to 1.9], Standard Error of Mean 0.78
Statistical Analysis 3: Comparison: PF-06372865 2.5 mg (Stage 1) vs PF-06372865 7.5 mg (Stage 1); [analysis description as in outcome 9, analysis 3]; Test type: Superiority or Other; p = 0.914, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.1, 90% CI 2-sided [-1.6 to 1.4], Standard Error of Mean 0.92
Statistical Analysis 4: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1); [analysis description as in outcome 9, analysis 4]; Test type: Superiority or Other; p = 0.892, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.1, 90% CI 2-sided [-1.3 to 1.5], Standard Error of Mean 0.86
Statistical Analysis 5: Comparison: Placebo (Stage 1) vs PF-06372865 2.5 mg (Stage 1); [analysis description as in outcome 9, analysis 5]; Test type: Superiority or Other; p = 0.463, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.6, 90% CI 2-sided [-0.8 to 2.0], Standard Error of Mean 0.82
Statistical Analysis 6: Comparison: PF-06372865 2.5 mg (Stage 1) vs PF-06372865 7.5 mg (Stage 1); [analysis description as in outcome 9, analysis 6]; Test type: Superiority or Other; p = 0.611, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.5, 90% CI 2-sided [-2.1 to 1.1], Standard Error of Mean 0.95
Statistical Analysis 7: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1); [analysis description as in outcome 9, analysis 7]; Test type: Superiority or Other; p = 0.321, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.9, 90% CI 2-sided [-0.6 to 2.4], Standard Error of Mean 0.88
Statistical Analysis 8: Comparison: Placebo (Stage 1) vs PF-06372865 2.5 mg (Stage 1); [analysis description as in outcome 9, analysis 8]; Test type: Superiority or Other; p = 0.294, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.9, 90% CI 2-sided [-0.5 to 2.3], Standard Error of Mean 0.85
Statistical Analysis 9: Comparison: PF-06372865 2.5 mg (Stage 1) vs PF-06372865 7.5 mg (Stage 1); [analysis description as in outcome 9, analysis 9]; Test type: Superiority or Other; p = 0.987, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.0, 90% CI 2-sided [-1.7 to 1.6], Standard Error of Mean 0.99
Statistical Analysis 10: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1); [analysis description as in outcome 9, analysis 10]; Test type: Superiority or Other; p = 0.599, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.5, 90% CI 2-sided [-1.2 to 2.3], Standard Error of Mean 1.04
Statistical Analysis 11: Comparison: Placebo (Stage 1) vs PF-06372865 2.5 mg (Stage 1); [analysis description as in outcome 9, analysis 11]; Test type: Superiority or Other; p = 0.322, Mixed-Effects Model Repeated Measure; LS Mean Difference = 1.0, 90% CI 2-sided [-0.7 to 2.6], Standard Error of Mean 1.0
Statistical Analysis 12: Comparison: PF-06372865 2.5 mg (Stage 1) vs PF-06372865 7.5 mg (Stage 1); [analysis description as in outcome 9, analysis 12]; Test type: Superiority or Other; p = 0.704, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.4, 90% CI 2-sided [-2.4 to 1.5], Standard Error of Mean 1.17
Statistical Analysis 13: Comparison: Placebo (Stage 2) vs PF-06372865 7.5 mg (Stage 2); [analysis description as in outcome 9, analysis 13]; Test type: Superiority or Other; p = 0.804, LS Mean Difference; LS Mean Difference = 0.3, 90% CI 2-sided [-2.0 to 2.7], Standard Error of Mean 1.38
Statistical Analysis 14: Comparison: Placebo (Stage 2) vs PF-06372865 2.5 mg (Stage 2); [analysis description as in outcome 9, analysis 14]; Test type: Superiority or Other; p = 0.559, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.8, 90% CI 2-sided [-3.2 to 1.6], Standard Error of Mean 1.38
Statistical Analysis 15: Comparison: PF-06372865 2.5 mg (Stage 2) vs PF-06372865 7.5 mg (Stage 2); [analysis description as in outcome 9, analysis 15]; Test type: Superiority or Other; p = 0.369, Mixed-Effects Model Repeated Measure; LS Mean Difference = 1.2, 90% CI 2-sided [-1.0 to 3.4], Standard Error of Mean 1.27
Statistical Analysis 16: Comparison: Placebo (Stage 2) vs PF-06372865 7.5 mg (Stage 2); [analysis description as in outcome 9, analysis 16]; Test type: Superiority or Other; p = 0.313, Mixed-Effects Model Repeated Measure; LS Mean Difference = 1.6, 90% CI 2-sided [-1.1 to 4.3], Standard Error of Mean 1.56
Statistical Analysis 17: Comparison: Placebo (Stage 2) vs PF-06372865 2.5 mg (Stage 2); [analysis description as in outcome 9, analysis 17]; Test type: Superiority or Other; p = 0.560, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.9, 90% CI 2-sided [-1.8 to 3.6], Standard Error of Mean 1.56
Statistical Analysis 18: Comparison: PF-06372865 2.5 mg (Stage 2) vs PF-06372865 7.5 mg (Stage 2); [analysis description as in outcome 9, analysis 18]; Test type: Superiority or Other; p = 0.635, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.7, 90% CI 2-sided [-1.8 to 3.2], Standard Error of Mean 1.43
Statistical Analysis 19: Comparison: Placebo (Stage 2) vs PF-06372865 7.5 mg (Stage 2); [analysis description as in outcome 9, analysis 19]; Test type: Superiority or Other; p = 0.538, Mixed-Effects Model Repeated Measure; LS Mean Difference = 1.0, 90% CI 2-sided [-1.8 to 3.8], Standard Error of Mean 1.62
Statistical Analysis 20: Comparison: Placebo (Stage 2) vs PF-06372865 2.5 mg (Stage 2); [analysis description as in outcome 9, analysis 20]; Test type: Superiority or Other; p = 0.942, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.1, 90% CI 2-sided [-2.7 to 2.9], Standard Error of Mean 1.60
Statistical Analysis 21: Comparison: PF-06372865 2.5 mg (Stage 2) vs PF-06372865 7.5 mg (Stage 2); [analysis description as in outcome 9, analysis 21]; Test type: Superiority or Other; p = 0.555, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.9, 90% CI 2-sided [-1.7 to 3.5], Standard Error of Mean 1.50
Statistical Analysis 22: Comparison: Placebo (Stage 2) vs PF-06372865 7.5 mg (Stage 2); [analysis description as in outcome 9, analysis 22]; Test type: Superiority or Other; p = 0.728, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.7, 90% CI 2-sided [-4.1 to 2.7], Standard Error of Mean 1.96
Statistical Analysis 23: Comparison: Placebo (Stage 2) vs PF-06372865 2.5 mg (Stage 2); [analysis description as in outcome 9, analysis 23]; Test type: Superiority or Other; p = 0.362, Mixed-Effects Model Repeated Measure; LS Mean Difference = -1.8, 90% CI 2-sided [-5.2 to 1.6], Standard Error of Mean 1.95
Statistical Analysis 24: Comparison: PF-06372865 2.5 mg (Stage 2) vs PF-06372865 7.5 mg (Stage 2); [analysis description as in outcome 9, analysis 24]; Test type: Superiority or Other; p = 0.538, Mixed-Effects Model Repeated Measure; LS Mean Difference = 1.1, 90% CI 2-sided [-2.0 to 4.3], Standard Error of Mean 1.81
Statistical Analysis 25: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1) vs Placebo (Stage 2) vs PF-06372865 7.5 mg (Stage 2); [analysis description as in outcome 13, analysis 25]; Test type: Superiority or Other; p = 0.949, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.1, 90% CI 2-sided [-2.0 to 1.8], Standard Error of Mean 1.11
Statistical Analysis 26: Comparison: Placebo (Stage 1) vs PF-06372865 2.5 mg (Stage 1) vs Placebo (Stage 2) vs PF-06372865 2.5 mg (Stage 2); [analysis description as in outcome 13, analysis 26]; Test type: Superiority or Other; p = 0.708, Mixed-Effects Model Repeated Measure; LS Mean Difference = -0.4, 90% CI 2-sided [-2.3 to 1.5], Standard Error of Mean 1.09
Statistical Analysis 27: Comparison: PF-06372865 2.5 mg (Stage 1) vs PF-06372865 7.5 mg (Stage 1) vs PF-06372865 2.5 mg (Stage 2) vs PF-06372865 7.5 mg (Stage 2); [analysis description as in outcome 13, analysis 27]; Test type: Superiority or Other; p = 0.752, Mixed-Effects Model Repeated Measure; LS Mean Difference = 0.3, 90% CI 2-sided [-1.5 to 2.2], Standard Error of Mean 1.07

15. Secondary Outcome: Percentage of Participants With Remission of Total Hamilton Anxiety Rating Scale (HAM-A) Scores
Description: Percentage of participants with HAM-A total score less than or equal to 7 in the last week of the Stage (Week 4 in Stage 1, Week 8 in Stage 2). The HAM-A scale was a clinician rated interview scale designed to measure the signs and symptoms of anxiety. It had 14-items to rate the intensity of psychic and somatic anxiety on a 5-point severity scale. Each item ranging from 0 (not present) to 4 (very severe) were summed up to give a total possible score of 0 (not present) to 56 (very severe), where lower scores indicates less anxiety.
Time Frame: Stage 1: Week 1 up to Week 4 and Stage 2: Week 5 up to Week 8
Population: Full analysis set for Stage 1 was defined as all participants randomized and who had received at least 1 dose of randomized treatment. The Stage 2 placebo non-responder set was defined as the subset of subjects in the Stage 2 placebo set who had both a <50% reduction in HAM-A between Stage 1 baseline and Week 4, and HAM-A value of >= 16 at Week 4.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Stage 1) | PF-06372865 2.5 mg (Stage 1) | PF-06372865 7.5 mg (Stage 1) | Placebo (Stage 2) | PF-06372865 2.5 mg (Stage 2) | PF-06372865 7.5 mg (Stage 2)
Number analyzed (Participants) | 45 | 24 | 21 | 6 | 8 | 8
percentage of participants | 6.67 | 12.50 | 4.76 | 0 | 0 | 12.50
Statistical Analysis 1: Comparison: Placebo (Stage 1) vs PF-06372865 7.5 mg (Stage 1); (PF-06372865 7.5 mg - Placebo). Logistic regression model includes treatment as fixed effect, and baseline as covariate. Baseline for Stage 1 is Day 1 and Stage 2 is Week 4 (Day 28); Test type: Superiority or Other; Regression, Logistic; Odds Ratio (OR) = 0.95, 90% CI 2-sided [0.37 to 2.45]
Statistical Analysis 2: Comparison: Placebo (Stage 1) vs PF-06372865 2.5 mg (Stage 1); (PF-06372865 2.5 mg - Placebo). Logistic regression model includes treatment as fixed effect, and baseline as covariate. Baseline for Stage 1 is Day 1 and Stage 2 is Week 4 (Day 28); Test type: Superiority or Other; Regression, Logistic; Odds Ratio (OR) = 1.64, 90% CI 2-sided [0.39 to 6.88]
Statistical Analysis 3: Comparison: PF-06372865 2.5 mg (Stage 1) vs PF-06372865 7.5 mg (Stage 1); (PF-06372865 7.5 mg - PF-06372865 2.5 mg). Logistic regression model includes treatment as fixed effect, and baseline as covariate. Baseline for Stage 1 is Day 1 and Stage 2 is Week 4 (Day 28); Test type: Superiority or Other; Regression, Logistic; Odds Ratio (OR) = 0.58, 90% CI 2-sided [0.23 to 1.49]

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and an serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non serious event during the study.
Groups:
- Placebo: All participants received placebo matched to PF-06372865 twice daily for 4 weeks in Stage 1 and Stage 2.
- PF-06372865 2.5 mg: All participants received PF-06372865 2.5 mg twice daily for 4 weeks in Stage 1 and Stage 2.
- PF-06372865 7.5 mg: All participants received PF-06372865 7.5 mg twice daily for 4 weeks in Stage 1 and Stage 2.
Arm/Group | Placebo | PF-06372865 2.5 mg | PF-06372865 7.5 mg
Serious Adverse Events (participants affected / at risk) | 1/87 | 0/37 | 0/35
Other Adverse Events (participants affected / at risk) | 27/87 | 13/37 | 16/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=87) | PF-06372865 2.5 mg (N=37) | PF-06372865 7.5 mg (N=35)
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=87) | PF-06372865 2.5 mg (N=37) | PF-06372865 7.5 mg (N=35)
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 2
Flatulence (Gastrointestinal disorders) | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 6 | 1 | 1
Fatigue (General disorders) | 4 | 2 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 2
Urinary tract infection (Infections and infestations) | 2 | 2 | 0
Dizziness (Nervous system disorders) | 5 | 1 | 7
Headache (Nervous system disorders) | 6 | 3 | 4
Somnolence (Nervous system disorders) | 5 | 3 | 5
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 2

LIMITATIONS AND CAVEATS:
All 34 centres who enrolled subjects were terminated due to internal sponsor portfolio prioritization. The decision to terminate the study was not due to any safety concern or change in the benefit:risk assessment of PF-06372865

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.